CLINICAL TRIAL: NCT01003691
Title: A PHASE 1, DOUBLE-MASKED, PLACEBO-CONTROLLED STUDY EVALUATING THE SAFETY, TOLERABILITY, IMMUNOGENICITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF MULTIPLE ESCALATING DOSAGES OF RN6G (PF-04382923) IN SUBJECTS WITH ADVANCED DRY, AGE-RELATED MACULAR DEGENERATION (AMD) INCLUDING GEOGRAPHIC ATROPHY
Brief Title: Safety And Tolerability Study Of RN6G In Subjects With Advanced Dry, Age-Related Macular Degeneration Including Geographic Atrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B1181002
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Age-Related Maculopathy; Age-Related Maculopathies; Eye Diseases; Retinal Degeneration; Macular Degeneration
Keywords: Phase 1b Advanced Dry Age-Related Macular Degeneration RN6G
MeSH Terms: conditions — Macular Degeneration; Eye Diseases; Retinal Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: RN6G; Biological: Placebo

INTERVENTIONS:
Biological: RN6G — Intravenous, multiple dose, dose ranging from 5 mg/kg up to a maximum of 15 mg/kg
Biological: Placebo — Intravenous, multiple dose with experimental dose

SUMMARY:
The purpose of this study is to determine the safety and tolerability of multiple doses of RN6G in subjects with advanced dry, age-related macular degeneration including geographic atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Be of non-child bearing potential
* Diagnosis of dry AMD including uni- or multi-focal geographic atrophy without foveal involvement
* BCVA of 20/50 or better in the study eye

Exclusion Criteria:

* Evidence of ocular disease other than advanced AMD or GA in the study eye
* History or diagnosis of exudative (wet) AMD, with subretinal or choroidal neovascular lesions in the study eye
* Presence of disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, central nervous immune, or gastrointestinal system
* Requires ocular or systemic medications that are known to be toxic to the lens, retina or optic nerve

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08-05 (Actual); Primary Completion 2013-03-05 (Actual); Study Completion 2013-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (24):
- United States (24):
  - Retinal Diagnostic Center, Campbell, California
  - American Institute of Research (Administrative Only), Los Gatos, California
  - Neurology Center Rai Kumar, San Jose, California
  - Harmeet Sachdev, MD, FAAN, San Jose, California
  - Santa Clara Drug, San Jose, California
  - Retina Associates of Florida, PA, Tampa, Florida
  - Hoye's Pharmacy, Tampa, Florida
  - Ranjit K. Sethi, MD, PC, Augusta, Georgia
  - Clinical Specialists, LLC, Augusta, Georgia
  - Southeast Retina Center, PC, Augusta, Georgia
  - University of Rochester Medical Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Hawthorne Pharmacy, West Columbia, South Carolina
  - Jay Markowitz and Associates, West Columbia, South Carolina
  - Palmetto Retina Center, LLC, West Columbia, South Carolina
  - South Carolina Neurological, West Columbia, South Carolina
  - National Central Pharmacy, Abilene, Texas
  - Abilene Surgery Center, Abilene, Texas
  - Heart and Vascular Institute, Abilene, Texas
  - Retina Research Institute of Texas, Abilene, Texas
  - Brian B. Berger, MD, PA, Austin, Texas
  - Retina Research Center, PLLC, Austin, Texas
  - Sleep Medicine Consultants, Austin, Texas
  - Specialty Compounding, Cedar Park, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1181002&StudyName=Safety%20And%20Tolerability%20Study%20Of%20RN6G%20In%20Subjects%20With%20Advanced%20Dry%2C%20Age-Related%20Macular%20Degeneration%20Including%20Geographic%20Atrophy

RESULTS

PARTICIPANT FLOW:
Groups:
- RN6G 5 mg/kg: RN6G (PF-04382923) 5 milligram/kilogram (mg/kg) of body weight, intravenous infusion over 60 minutes every 4 weeks until unacceptable toxicity, up to Month 5.
- RN6G 10 mg/kg: RN6G (PF-04382923) 10 mg/kg of body weight, intravenous infusion over 60 minutes every 4 weeks until unacceptable toxicity, up to Month 5.
- RN6G 15 mg/kg: RN6G (PF-04382923) 15 mg/kg of body weight, intravenous infusion over 60 minutes every 4 weeks until unacceptable toxicity, up to Month 5.
- Placebo: Placebo intravenous infusion over 60 minutes, every 4 weeks, until unacceptable toxicity, up to Month 5.
Period: Overall Study
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Customized [Count of Participants; unit: Participants]
  60 to less than (<) 75 years | 3 | 3 | 3 | 2 | 11
  Greater than or equal to (>=) 75 years | 3 | 3 | 3 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5 | 3 | 13
  Male | 2 | 5 | 1 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 6 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 5 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Toxicity or Intolerable Dose Criteria
Description: The dose was considered intolerable if a participant developed either ocular toxicity or other toxicity as per Common Terminology Criteria for Adverse Events (CTCAE) or based on the investigator's discretion. Ocular toxicity included: Grade >= 3 (retinopathy, retinal detachment, cataract formation, optic disk edema, keratitis, vitreous hemorrhage and uveitis) and acute vision loss of greater than 3 lines of vision up to and including 140 days after the first dose. Other toxicity included serious adverse event (SAE), Grade >= 3 (increased liver transaminases, encephalopathy/leukoencephalopathy, diarrhea, enteritis or nausea, prolongation of QT interval [Fridericia's correction]), Grade >=2 (central nervous system hemorrhage, decreased total leukocyte count, increased serum creatinine) and thrombocytopenia <100*10 9 /liter.
Time Frame: Baseline up to Day 304/End of Treatment (ET)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug or placebo.
Measure: Number; unit: Participants
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Categorized by Severity
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to Day 304/ET that were absent before treatment or that worsened relative to pretreatment state. AE was assessed according to severity; Grade 1 (mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated), Grade 2 (moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living [ADL]), Grade 3 (severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL), Grade 4 (life-threatening consequences; urgent intervention indicated) and Grade 5 (death related to AE).
Time Frame: Baseline up to Day 304/ET
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Grade 1 | 1 | 3 | 0 | 0
  Grade 2 | 5 | 3 | 4 | 5
  Grade 3 | 0 | 0 | 2 | 1
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): All Causalities and TEAEs Categorized by Causal Relationship to Study Drug
Description: All causalities AE was any untoward medical occurrence in participant who received study drug without regard to causal relationship. Drug-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to Day 304/ET that were absent before treatment or that worsened relative to pretreatment state. All causalities and drug-related AEs reported wherein drug-related AEs were reported as ocular and non-ocular AEs. Ocular AEs were events which were localized in the ocular region and non-ocular AEs were systemic events which were not localized but occurred throughout the systemic circulation.
Time Frame: Baseline up to Day 304/ET
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  All causalities AE | 6 | 6 | 6 | 6
  Drug-related Ocular AE | 0 | 0 | 0 | 0
  Drug-related non-ocular AE | 2 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Ocular Treatment Emergent Adverse Events (TEAEs) Categorized by Severity
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to Day 304/ET that were absent before treatment or that worsened relative to pretreatment state. Ocular AE were events which were localized in the ocular region and was assessed according to severity; Grade 1 (mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated), Grade 2 (moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL), Grade 3 (severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL), Grade 4 (life-threatening consequences; urgent intervention indicated) and Grade 5 (death related to AE).
Time Frame: Baseline up to Day 304/ET
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Grade 1 | 4 | 4 | 0 | 2
  Grade 2 | 0 | 0 | 3 | 2
  Grade 3 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Ocular Treatment Emergent Adverse Events (TEAEs) Categorized by Causal Relationship to Study Drug
Description: AE was any untoward medical occurrence in participant who received study drug without regard to causal relationship and drug-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to Day 304/ET that were absent before treatment or that worsened relative to pretreatment state. Ocular AEs were events which were localized in the ocular region. Ocular AEs reported as related and non-related to study drug.
Time Frame: Baseline up to Day 304/ET
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Related | 0 | 0 | 0 | 0
  Not Related | 4 | 4 | 3 | 4

6. Primary Outcome: Number of Participants With Systemic Treatment Emergent Adverse Events (TEAEs) Categorized by Severity
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to Day 304/ET that were absent before treatment or that worsened relative to pretreatment state. Systemic AE were events which were not localized but occurred throughout the systemic circulation and was assessed according to severity; Grade 1 (mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated), Grade 2 (moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL), Grade 3 (severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL), Grade 4 (life-threatening consequences; urgent intervention indicated) and Grade 5 (death related to AE).
Time Frame: Baseline up to Day 304/ET
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Grade 1 | 1 | 3 | 0 | 0
  Grade 2 | 5 | 3 | 4 | 5
  Grade 3 | 0 | 0 | 2 | 1
  Grade 4 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Systemic Treatment Emergent Adverse Events (TEAEs) Categorized by Causal Relationship to Study Drug
Description: AE was any untoward medical occurrence in participant who received study drug without regard to causal relationship and drug-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to Day 304/ET that were absent before treatment or that worsened relative to pretreatment state. Systemic TEAEs were events which were not localized but occurred throughout the systemic circulation and reported as related and non-related to study drug.
Time Frame: Baseline up to Day 304/ET
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Related | 2 | 0 | 0 | 0
  Not related | 4 | 6 | 6 | 6

8. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of RN6G (PF-04382923)
Description: Area under the concentration-time profile from time zero to time tau (τ), the dosing interval, where tau = 672 hours.
Time Frame: Pre-dose: 0 hour on Day 1, 28, 56, 84,112,140; Post-dose: 1, 2, 4, 24, 168, 336 hours on Day 1 and 1, 2, 4, 24, 336, 672 hours on Day 140
Population: Analysis population included all randomized participants who met the inclusion criteria and received any amount of study drug. Here "Overall Number of participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluated for specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour per milliliter (mcg*h/mL)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
Microgram*hour per milliliter (mcg*h/mL)
  Day 1: number analyzed (Participants) | 2 | 0 | 2
  Day 1 | NA (NA) — Data for geometric mean and geometric CV not estimable as only 2 participants were evaluated, individual values were 18800 and 21200 mcg*h/mL |  | NA (NA) — Data for geometric mean and geometric CV not estimable as only 2 participants were evaluated, individual values were 73500 and 80000 mcg*h/mL
  Day 140 | 50230 (20) | 140300 (14) | 213200 (16)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of RN6G (PF-04382923)
Time Frame: Pre-dose: 0 hour on Day 1, 28, 56, 84,112,140; Post-dose: 1, 2, 4, 24, 168, 336 hours on Day 1 and 1, 2, 4, 24, 336, 672, 1992, 3936 hours on Day 140
Population: All randomized participants who met the inclusion criteria and received any amount of study drug were included. Here "Overall Number of participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
Microgram per milliliter (mcg/mL)
  Day 1 | 142.9 (12) | 283.4 (18) | 524.1 (66)
  Day 140 | 185.1 (16) | 439.8 (15) | 691.7 (12)

10. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of RN6G (PF-04382923)
Time Frame: Pre-dose: 0 hour on Day 1, 28, 56, 84,112,140; Post-dose: 1, 2, 4, 24, 336, 672, 1992, 3936 hours on Day 140
Population: Analysis population included all randomized participants who met the inclusion criteria and received any amount of study drug. Here "Overall Number of participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
Microgram per milliliter (mcg/mL) | 38.43 (40) | 119.7 (23) | 201.5 (27)

11. Secondary Outcome: Plasma Concentration (Css) at Steady State of RN6G (PF-04382923)
Description: Css is the concentration of the drug at the state when the amount of drug administered is equal to the amount of drug eliminated.
Time Frame: Pre-dose: 0 hour on Day 1, 28, 56, 84,112,140; Post-dose: 1, 2, 4, 24, 336, 672, 1992, 3936 hours on Day 140
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
Microgram per milliliter (mcg/mL) | 74.75 (20) | 208.7 (14) | 317.2 (16)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of RN6G (PF-04382923)
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Median (Full Range); unit: Hour
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
Hour
  Day 1 | 1.49 [1.00 to 3.00] | 2.06 [1.17 to 4.08] | 2.17 [1.03 to 4.98]
  Day 140 | 1.77 [1.02 to 2.13] | 2.05 [1.00 to 5.30] | 1.32 [1.03 to 1.33]

13. Secondary Outcome: Volume of Distribution at Steady State (Vss) of RN6G (PF-04382923)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: Pre-dose: 0 hour on Day 1, 28, 56, 84,112,140; Post-dose: 1, 2, 4, 24, 336, 672, 1992, 3936 hours on Day 140
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per kilogram (mL/kg)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
Milliliter per kilogram (mL/kg) | 79.52 (23) | 88.04 (26) | 78.45 (11)

14. Secondary Outcome: Mean Residence Time (MRT) of RN6G (PF-04382923)
Description: The mean total time drug resides in the body.
Time Frame: Pre-dose: 0 hour on Day 1, 28, 56, 84,112,140; Post-dose: 1, 2, 4, 24, 336, 672, 1992, 3936 hours on Day 140
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
Hour | 818.1 (182.15) | 1274 (352.28) | 1121 (135.38)

15. Secondary Outcome: Systemic Clearance (CL) of RN6G (PF-04382923)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Pre-dose: 0 hour on Day 1, 28, 56, 84,112,140; Post-dose: 1, 2, 4, 24, 336, 672, 1992, 3936 hours on Day 140
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour per kilogram
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
Milliliter per hour per kilogram | 0.09954 (20) | 0.07129 (14) | 0.07036 (16)

16. Secondary Outcome: Plasma Decay Half-Life (t1/2) of RN6G (PF-04382923)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose: 0 hour on Day 1, 28, 56, 84,112,140; Post-dose: 1, 2, 4, 24, 336, 672, 1992, 3936 hours on Day 140
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg
Number analyzed (Participants) | 6 | 6 | 5
Hour | 25.14 (5.0774) | 42.00 (6.6321) | 38.10 (4.9738)

17. Secondary Outcome: Change From Baseline in Plasma Total Amyloid (A) Beta (1-X) Concentration at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET
Description: Amyloid (A) Beta (1-X) is a primary activator of complement in Alzheimer's disease (AD).
Time Frame: Baseline, Day 1 (1 hour, 2 hours, 4 hours post dose), 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140 (predose, 1 hour, 2 hours, 4 hours post dose), 141, 154, 168, 224, 304/ET
Population: All randomized participants who met the inclusion criteria and received any amount of study drug were included. Here "Number Analyzed" signifies number of participants evaluated for given time point.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter (pg/ml)
Groups:
- Placebo: Placebo matching to PF-04382923 in dosages ranging from 5 to 15 mg/kg as intravenous infusion over 60 minutes followed by a 5 mL flush of 0.9% Sodium Chloride Injection, every 4 weeks, for a total of up to 6 doses.
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Picogram per milliliter (pg/ml)
  Baseline: number analyzed (Participants) | 6 | 6 | 5 | 6
  Baseline | 371.8 (284.73) | 1596.8 (2794.08) | 200.0 (0.00) | 386.5 (174.33)
  Change at 1H post-dose Day 1: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at 1H post-dose Day 1 | 3340.5 (386.71) | 3205.5 (856.06) | 3947.2 (1822.39) | 0.3 (83.39)
  Change at 2H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 5 | 6
  Change at 2H post-dose Day 1 | 5118.7 (709.00) | 4821.2 (1114.32) | 5610.8 (2544.70) | 45.3 (125.22)
  Change at 4H post-dose Day 1: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at 4H post-dose Day 1 | 7850.0 (1490.33) | 6992.7 (1716.83) | 7874.3 (2158.56) | 1.7 (225.19)
  Change at Day 2: number analyzed (Participants) | 6 | 4 | 4 | 6
  Change at Day 2 | 33804.2 (5420.83) | 33566.0 (4698.42) | 37862.0 (1069.86) | -9.8 (132.42)
  Change at Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 7 | 50329.3 (9389.75) | 88678.7 (22431.39) | 94017.0 (7060.55) | 16.8 (52.82)
  Change at Day 14: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 14 | 25303.0 (4293.92) | 69611.3 (21077.31) | 80138.0 (13795.55) | -66.2 (103.72)
  Change at Day 19: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 19 | 17782.7 (4264.51) | 54407.7 (15467.03) | 71190.6 (7553.42) | -62.5 (106.16)
  Change at Day 28: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 28 | 8777.5 (1441.65) | 35848.3 (9540.26) | 57701.0 (14705.10) | -69.7 (239.14)
  Change at Day 45: number analyzed (Participants) | 6 | 5 | 5 | 6
  Change at Day 45 | 41329.3 (12376.68) | 87735.4 (19304.46) | 110278.0 (20296.92) | -6.5 (209.72)
  Change at Day 56: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 56 | 23723.0 (4080.35) | 70846.5 (24378.68) | 98343.8 (21336.44) | -36.3 (305.27)
  Change at Day 75: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 75 | 42393.7 (7739.27) | 121176.2 (34652.27) | 149272.0 (23898.10) | 205.6 (302.40)
  Change at Day 84: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 84 | 29386.3 (3246.30) | 89908.2 (28896.82) | 120091.6 (5895.10) | 122.2 (362.01)
  Change at Day 103: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 103 | 50269.8 (7129.73) | 114474.3 (28268.90) | 157448.0 (33235.41) | 116.6 (296.52)
  Change at Day 112: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112 | 34071.5 (4062.24) | 107243.5 (28813.61) | 140917.6 (17498.78) | 214.4 (342.45)
  Change at Day 131: number analyzed (Participants) | 5 | 6 | 4 | 5
  Change at Day 131 | 62226.8 (17554.96) | 124417.0 (26689.05) | 168767.8 (7272.93) | -61.6 (131.01)
  Change at pre-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at pre-dose Day 140 | 46295.7 (7585.69) | 102548.2 (22902.22) | 154350.0 (9459.75) | -3.4 (92.42)
  Change at 1 H post-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 1 H post-dose Day 140 | 41991.0 (7209.04) | 98349.2 (20226.44) | 140246.0 (15770.21) | -25.0 (80.53)
  Change at 2 H Post-dose Day 140: number analyzed (Participants) | 6 | 6 | 4 | 4
  Change at 2 H Post-dose Day 140 | 49017.8 (6793.71) | 102384.7 (17624.73) | 136109.5 (12883.65) | -137.3 (135.93)
  Change at 4 H Post-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 4 H Post-dose Day 140 | 51102.8 (6552.83) | 101938.3 (21440.86) | 153793.0 (15312.09) | -144.2 (158.04)
  Change at Day 141: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 141 | 27212.1 (12018.62) | 36042.0 (25934.30) | 80464.2 (11546.49) | -11.0 (30.66)
  Change at Day 154: number analyzed (Participants) | 0 | 6 | 5 | 4
  Change at Day 154 |  | 141033.8 (22685.63) | 190913.6 (29331.01) | -103.5 (85.83)
  Change at Day 168: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 168 | 52558.0 (6374.13) | 103651.8 (27880.97) | 161691.4 (21292.74) | -64.6 (132.40)
  Change at Day 224: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 224 | 20950.3 (6951.30) | 35489.0 (11571.26) | 57692.0 (16310.16) | -110.3 (138.97)
  Change at day 304/ET: number analyzed (Participants) | 0 | 6 | 5 | 4
  Change at day 304/ET |  | 13550.8 (5901.76) | 12127.2 (3196.16) | -164.3 (167.57)

18. Secondary Outcome: Percent Change From Baseline in Plasma Total Amyloid (A) Beta (1-X) Concentration at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET
Time Frame: Day 1 (1 hour , 2 hours, 4 hours post dose), 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140 (predose, 1 hour, 2 hours, 4 hours post dose), 141, 154, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percent change
  Percent change at 1 H post-dose Day 1: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at 1 H post-dose Day 1 | 1194.4 (541.02) | 1032.9 (860.01) | 1973.6 (911.19) | 3.8 (21.25)
  Percent change at 2 H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 5 | 6
  Percent change at 2 H post-dose Day 1 | 1835.9 (859.97) | 1682.9 (1332.55) | 2805.4 (1272.35) | 17.7 (37.96)
  Percentage change at 4 H post-dose Day 1: number analyzed (Participants) | 6 | 6 | 4 | 6
  Percentage change at 4 H post-dose Day 1 | 2899.5 (1575.11) | 2044.5 (1595.93) | 3937.1 (1079.28) | 14.5 (61.22)
  Percent change at Day 2: number analyzed (Participants) | 6 | 4 | 4 | 6
  Percent change at Day 2 | 11999.3 (5344.01) | 9771.3 (6115.66) | 18931.0 (534.93) | 4.3 (29.32)
  Percent change at Day 7: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 7 | 17643.7 (7989.43) | 22214.1 (16132.62) | 47008.5 (3530.28) | 3.1 (13.89)
  Percent change at Day 14: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 14 | 8930.3 (3978.36) | 16692.0 (11490.17) | 40069.0 (6897.78) | -12.4 (20.10)
  Percent change at Day 19: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 19 | 6096.9 (2660.58) | 13136.7 (9098.67) | 35595.3 (3776.71) | -13.2 (18.08)
  Percent change at Day 28: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 28 | 3168.7 (1297.49) | 8714.5 (5831.88) | 28850.5 (7352.55) | -3.3 (72.57)
  Percent change at Day 45: number analyzed (Participants) | 6 | 5 | 5 | 6
  Percent change at Day 45 | 14458.4 (7747.84) | 25626.3 (16350.32) | 55139.0 (10148.46) | 19.0 (84.63)
  Percent change at Day 56: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 56 | 8156.5 (3005.78) | 16396.4 (11269.80) | 49171.9 (10668.22) | 20.9 (120.63)
  Percent change at Day 75: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 75 | 14815.6 (6477.51) | 29483.6 (20874.07) | 74636.0 (11949.05) | 72.3 (122.02)
  Percent change at Day 84: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 84 | 10497.3 (4494.06) | 21128.7 (14305.48) | 60045.8 (2947.55) | 51.2 (124.25)
  Percent change at Day 103: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 103 | 17482.8 (6740.53) | 28726.4 (20620.23) | 78724.0 (16617.70) | 48.2 (120.26)
  Percent change at Day 112: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 112 | 12401.6 (5938.63) | 26653.1 (19128.49) | 70458.8 (8749.39) | 75.8 (138.85)
  Percent change at Day 131: number analyzed (Participants) | 5 | 6 | 4 | 5
  Percent change at Day 131 | 20902.9 (8509.92) | 31839.9 (22850.11) | 84383.9 (3636.46) | -6.5 (28.29)
  Percent change at Pre-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Pre-dose Day 140 | 16323.4 (6890.74) | 26584.4 (19667.93) | 77175.0 (4729.87) | 6.8 (25.29)
  Percent change at 1 H Post dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at 1 H Post dose Day 140 | 15067.2 (6922.60) | 25462.2 (18562.61) | 70123.0 (7885.10) | -2.3 (23.04)
  Percent change at 2 H Post dose Day 140: number analyzed (Participants) | 6 | 6 | 4 | 4
  Percent change at 2 H Post dose Day 140 | 17418.4 (7204.24) | 27192.5 (19768.55) | 68054.8 (6441.82) | -25.9 (21.26)
  Percent change at 4 H Post dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at 4 H Post dose Day 140 | 18171.1 (7481.91) | 26342.6 (19070.40) | 76896.5 (7656.04) | -29.4 (24.61)
  Percent change at Day 141: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 141 | 27212.1 (12018.62) | 36042.0 (25934.30) | 80464.2 (11546.49) | -11.0 (30.66)
  Percent change at Day 154: number analyzed (Participants) | 0 | 6 | 5 | 4
  Percent change at Day 154 |  | 37731.7 (28276.18) | 95456.8 (14665.51) | -21.2 (14.56)
  Percent change at Day 168: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 168 | 19415.4 (9203.47) | 26639.1 (19545.03) | 80845.7 (10646.37) | -10.1 (29.15)
  Percent change at Day 224: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 224 | 7954.0 (5003.96) | 9003.9 (7319.06) | 28846.0 (8155.08) | -22.2 (27.76)
  Percent change at Day 304 / ET: number analyzed (Participants) | 0 | 6 | 5 | 4
  Percent change at Day 304 / ET |  | 3182.9 (2499.39) | 6063.6 (1598.08) | -31.6 (27.03)

19. Secondary Outcome: Change From Baseline in Plasma Amyloid (A) Beta (1-40) Concentration at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET
Time Frame: Baseline, Day 1 (1 hour , 2 hours, 4 hours post dose), 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140 (predose, 1 hour, 2 hours, 4 hours post dose), 141, 154, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Picogram per milliliter (pg/ml)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Picogram per milliliter (pg/ml)
  Baseline: number analyzed (Participants) | 6 | 6 | 5 | 6
  Baseline | 160.4 (36.33) | 199.7 (24.19) | 209.2 (13.26) | 224.3 (61.26)
  Change at 1H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 5 | 6
  Change at 1H post-dose Day 1 | 1271.3 (131.35) | 1306.4 (184.77) | 1548.8 (398.99) | -3.7 (21.10)
  Change at 2 H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 4 | 6
  Change at 2 H post-dose Day 1 | 1939.6 (185.16) | 2082.4 (457.09) | 2264.8 (438.40) | -0.7 (27.10)
  Change at 4 H post-dose Day 1: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at 4 H post-dose Day 1 | 3159.6 (510.52) | 3290.3 (525.32) | 3202.3 (730.89) | 4.2 (27.80)
  Change at Day 2: number analyzed (Participants) | 6 | 4 | 4 | 6
  Change at Day 2 | 10071.3 (1097.81) | 10256.8 (1125.20) | 11164.8 (563.89) | -5.5 (21.94)
  Change at Day 7: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 7 | 12089.6 (2224.22) | 18817.0 (4600.38) | 24150.8 (3178.81) | -2.8 (16.02)
  Change at Day 14: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 14 | 6047.9 (751.77) | 16450.3 (4571.75) | 19050.8 (3495.78) | -6.5 (13.91)
  Change at Day 19: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 19 | 4626.3 (506.10) | 12467.0 (3360.84) | 17990.8 (4568.62) | 8.2 (27.46)
  Change at Day 28: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 28 | 2809.6 (534.82) | 9117.0 (2492.73) | 15410.8 (3844.36) | -3.0 (17.44)
  Change at Day 45: number analyzed (Participants) | 6 | 5 | 5 | 6
  Change at Day 45 | 10302.9 (2886.26) | 18746.0 (4221.27) | 24150.8 (1138.42) | -7.7 (46.88)
  Change at Day 56: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 56 | 6352.9 (513.41) | 14645.3 (5174.94) | 20630.8 (3400.87) | -16.8 (46.67)
  Change at Day 75: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 75 | 10751.3 (796.75) | 24750.3 (5951.71) | 26910.8 (1110.60) | -33.0 (24.37)
  Change at Day 84: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 84 | 7687.9 (915.03) | 20800.3 (6538.53) | 23270.8 (1691.32) | -15.6 (61.32)
  Change at Day 103: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 103 | 12239.6 (1315.07) | 25900.3 (6385.93) | 29170.8 (5936.75) | -15.6 (36.92)
  Change at Day 112: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112 | 8517.9 (1608.78) | 23517.0 (6359.32) | 28250.8 (2534.65) | -18.6 (35.53)
  Change at Day 131: number analyzed (Participants) | 6 | 6 | 4 | 5
  Change at Day 131 | 15272.9 (2939.43) | 26550.3 (5860.63) | 37614.8 (8703.34) | 7.0 (56.04)
  Change at pre-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at pre-dose Day 140 | 10402.9 (1699.34) | 20192.0 (10768.73) | 33910.8 (4820.26) | 26.8 (102.19)
  Change at 1 H post-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 1 H post-dose Day 140 | 12626.3 (2294.39) | 25550.3 (6073.42) | 34470.8 (7089.10) | -9.0 (41.35)
  Change at 2 H Post-dose Day 140: number analyzed (Participants) | 6 | 6 | 4 | 4
  Change at 2 H Post-dose Day 140 | 13922.9 (2470.45) | 26717.0 (5581.26) | 36114.8 (6268.68) | -31.0 (27.60)
  Change at 4 H Post-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 4 H Post-dose Day 140 | 15889.6 (1923.62) | 25283.7 (5234.95) | 36750.8 (14910.47) | -27.4 (38.63)
  Change at Day 141: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 141 | 20889.6 (2456.19) | 31733.7 (6395.71) | 39990.8 (8261.80) | -24.2 (40.38)
  Change at Day 154: number analyzed (Participants) | 0 | 6 | 5 | 4
  Change at Day 154 |  | 25050.3 (5480.90) | 47310.8 (2244.59) | -35.8 (37.98)
  Change at Day 168: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 168 | 11557.9 (2152.82) | 21517.0 (5926.14) | 36750.8 (5023.07) | -20.4 (52.83)
  Change at Day 224: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 224 | 3534.6 (1383.04) | 8518.7 (2946.68) | 14190.8 (3337.13) | 15.3 (66.79)
  Change at day 304/ET: number analyzed (Participants) | 0 | 6 | 5 | 4
  Change at day 304/ET |  | 2483.7 (1124.28) | 3340.8 (994.48) | 26.8 (87.01)

20. Secondary Outcome: Percent Change From Baseline in Plasma Amyloid (A) Beta (1-40) Concentrations at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET
Time Frame: Day 1 (1 hour, 2 hours, 4 hours post dose), 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140 (predose, 1 hour, 2 hours, 4 hours post dose), 141, 154, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
percent change
  Percent change at 1 H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 5 | 6
  Percent change at 1 H post-dose Day 1 | 838.8 (262.62) | 660.9 (101.20) | 752.8 (247.20) | 0.4 (9.79)
  Percent change at 2 H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 4 | 6
  Percent change at 2 H post-dose Day 1 | 1283.4 (428.98) | 1051.5 (230.65) | 1082.6 (225.11) | 1.8 (12.92)
  Percent change at 4 H post-dose Day 1: number analyzed (Participants) | 6 | 6 | 4 | 6
  Percent change at 4 H post-dose Day 1 | 2129.1 (971.74) | 1649.8 (190.06) | 1509.3 (255.86) | 3.2 (12.13)
  Percent change at Day 2: number analyzed (Participants) | 6 | 4 | 4 | 6
  Percent change at Day 2 | 6536.9 (1533.60) | 5332.4 (437.02) | 5328.4 (422.35) | -0.4 (10.07)
  Percent change at Day 7: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 7 | 8153.4 (3691.20) | 9483.1 (2136.77) | 11658.5 (2346.26) | -1.0 (7.54)
  Percent change at Day 14: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 14 | 4001.5 (1313.42) | 8124.3 (1400.09) | 9132.2 (1770.33) | -2.1 (5.38)
  Percent change at Day 19: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 19 | 3048.1 (934.03) | 6169.0 (996.40) | 8606.3 (2099.47) | 6.5 (15.76)
  Percent change at Day 28: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 28 | 1836.7 (528.74) | 4501.8 (758.64) | 7485.9 (2422.75) | -0.7 (8.35)
  Percent change at Day 45: number analyzed (Participants) | 6 | 5 | 5 | 6
  Percent change at Day 45 | 6632.8 (2095.25) | 9614.6 (1371.10) | 11600.4 (1173.09) | 1.0 (22.07)
  Percent change at Day 56: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 56 | 4104.0 (781.38) | 7229.3 (1982.40) | 9938.9 (2032.57) | -2.8 (23.72)
  Percent change at Day 75: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 75 | 7033.1 (1783.12) | 12296.0 (1777.75) | 12933.0 (1384.70) | -12.5 (9.43)
  Percent change at Day 84: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 84 | 5034.2 (1396.44) | 10287.0 (2294.92) | 11153.8 (978.44) | -3.5 (28.74)
  Percent change at Day 103: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 103 | 8033.3 (2202.15) | 12858.0 (1914.67) | 14043.1 (3217.61) | -4.5 (16.16)
  Percent change at Day 112: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 112 | 5736.6 (2367.32) | 11719.8 (2354.18) | 13528.7 (1209.21) | -6.4 (15.20)
  Percent change at Day 131: number analyzed (Participants) | 6 | 6 | 4 | 5
  Percent change at Day 131 | 9742.8 (1628.75) | 13197.8 (1567.68) | 17840.0 (3578.16) | 4.9 (23.25)
  Percent change at Pre-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Pre-dose Day 140 | 6750.1 (1605.57) | 9991.6 (4745.47) | 16216.1 (2105.17) | 16.6 (51.02)
  Percent change at 1 H Post dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at 1 H Post dose Day 140 | 8274.4 (2373.14) | 12713.5 (2035.10) | 16473.9 (3063.74) | -1.5 (18.15)
  Percent change at 2 H Post dose Day 140: number analyzed (Participants) | 6 | 6 | 4 | 4
  Percent change at 2 H Post dose Day 140 | 9035.4 (2212.53) | 13326.7 (1838.41) | 17173.8 (2625.79) | -11.2 (9.09)
  Percent change at 4 H Post dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at 4 H Post dose Day 140 | 10332.3 (2454.30) | 12606.4 (1626.29) | 17656.9 (7083.30) | -9.6 (13.47)
  Percent change at Day 141: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 141 | 13778.6 (4413.73) | 15838.7 (2208.15) | 19190.4 (4117.80) | -7.8 (15.61)
  Percent change at Day 154: number analyzed (Participants) | 0 | 6 | 5 | 4
  Percent change at Day 154 |  | 12461.9 (1481.16) | 22722.9 (2317.53) | -12.7 (13.89)
  Percent change at Day 168: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 168 | 7539.0 (2097.66) | 10766.1 (2561.52) | 17703.0 (3291.42) | -5.3 (22.33)
  Percent change at Day 224: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 224 | 2277.4 (870.42) | 4228.9 (1141.96) | 6880.8 (2087.34) | 14.5 (35.70)
  Percent change at Day 304 / ET: number analyzed (Participants) | 0 | 6 | 5 | 4
  Percent change at Day 304 / ET |  | 1263.2 (640.49) | 1603.7 (481.43) | 10.9 (32.02)

21. Secondary Outcome: Change From Baseline in Plasma Amyloid (A) Beta (1-42) Concentration at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/ml)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
picogram per milliliter (pg/ml)
  Baseline: number analyzed (Participants) | 6 | 6 | 5 | 6
  Baseline | 34.0 (5.61) | 67.3 (36.14) | 46.9 (8.62) | 61.4 (31.71)
  Change at 1H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 5 | 6
  Change at 1H post-dose Day 1 | 65.3 (15.08) | 72.4 (14.51) | 154.9 (49.51) | -7.7 (16.71)
  Change at 2 H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 4 | 6
  Change at 2 H post-dose Day 1 | 84.6 (21.50) | 126.8 (36.79) | 193.9 (65.55) | -4.0 (19.86)
  Change at 4 H post-dose Day 1: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at 4 H post-dose Day 1 | 100.0 (18.50) | 179.5 (34.06) | 262.6 (113.24) | 4.0 (5.75)
  Change at Day 2: number analyzed (Participants) | 6 | 4 | 4 | 6
  Change at Day 2 | 88.6 (32.58) | 194.8 (48.89) | 328.4 (99.74) | -13.3 (26.69)
  Change at Day 7: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 7 | 42.1 (16.79) | 77.4 (26.92) | 144.1 (35.08) | 3.9 (32.00)
  Change at Day 14: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 14 | 18.7 (9.18) | 42.4 (43.12) | 75.9 (19.03) | 9.1 (22.03)
  Change at Day 19: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 19 | 13.9 (5.23) | 33.2 (34.62) | 71.2 (13.06) | 8.4 (22.71)
  Change at Day 28: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 28 | 4.8 (3.31) | 8.4 (28.46) | 68.3 (29.29) | -4.3 (11.73)
  Change at Day 45: number analyzed (Participants) | 6 | 5 | 5 | 6
  Change at Day 45 | 31.3 (7.24) | 50.9 (31.77) | 123.1 (23.36) | -12.6 (25.16)
  Change at Day 56: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 56 | 18.0 (7.94) | 56.6 (61.02) | 101.3 (25.80) | -15.9 (28.84)
  Change at Day 75: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 75 | 28.9 (11.25) | 78.0 (51.53) | 144.5 (29.38) | -22.3 (27.87)
  Change at Day 84: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 84 | 25.6 (3.60) | 56.3 (54.71) | 104.1 (21.92) | -14.7 (26.98)
  Change at Day 103: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 103 | 41.9 (6.37) | 94.4 (49.79) | 141.1 (47.02) | -17.8 (28.09)
  Change at Day 112: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112 | 26.2 (8.53) | 88.2 (58.68) | 124.9 (39.52) | -18.8 (22.91)
  Change at Day 131: number analyzed (Participants) | 6 | 6 | 4 | 5
  Change at Day 131 | 56.3 (11.71) | 115.0 (68.50) | 180.1 (18.23) | -19.9 (24.25)
  Change at pre-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at pre-dose Day 140 | 37.2 (8.51) | 80.2 (59.94) | 136.3 (9.43) | -10.9 (43.12)
  Change at 1 H post-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 1 H post-dose Day 140 | 87.8 (10.70) | 177.5 (67.55) | 257.7 (63.99) | -21.7 (25.89)
  Change at 2 H Post-dose Day 140: number analyzed (Participants) | 6 | 6 | 4 | 4
  Change at 2 H Post-dose Day 140 | 113.2 (19.82) | 209.2 (51.64) | 292.9 (57.03) | -28.7 (31.64)
  Change at 4 H Post-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 4 H Post-dose Day 140 | 132.3 (12.73) | 243.7 (58.08) | 360.9 (66.62) | -10.5 (39.49)
  Change at Day 141: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 141 | 120.0 (15.08) | 280.2 (81.80) | 404.7 (84.86) | -26.1 (24.22)
  Change at Day 154: number analyzed (Participants) | 0 | 6 | 5 | 4
  Change at Day 154 |  | 113.4 (72.67) | 229.5 (29.57) | -29.3 (25.98)
  Change at Day 168: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 168 | 39.5 (4.78) | 72.7 (50.70) | 168.9 (34.85) | -21.9 (27.63)
  Change at Day 224: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 224 | 8.6 (9.82) | -1.8 (41.26) | 45.6 (14.60) | -8.5 (42.38)
  Change at day 304/ET: number analyzed (Participants) | 0 | 6 | 5 | 3
  Change at day 304/ET |  | -3.6 (40.36) | 4.8 (5.31) | -35.9 (26.66)

22. Secondary Outcome: Percent Change From Baseline in Plasma Amyloid (A) Beta (1-42) Concentrations at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET
Time Frame: as for outcome 20
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
percent change
  Percent change at 1 H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 5 | 6
  Percent change at 1 H post-dose Day 1 | 199.0 (74.28) | 163.7 (102.35) | 340.2 (133.10) | -7.0 (20.63)
  Percent change at 2 H post-dose Day 1: number analyzed (Participants) | 6 | 5 | 4 | 6
  Percent change at 2 H post-dose Day 1 | 257.8 (101.75) | 254.3 (104.05) | 412.7 (98.90) | 0.5 (23.12)
  Percent change at 4 H post-dose Day 1: number analyzed (Participants) | 6 | 6 | 4 | 6
  Percent change at 4 H post-dose Day 1 | 306.4 (111.88) | 341.8 (174.55) | 545.8 (131.45) | 10.4 (12.86)
  Percent change at Day 2: number analyzed (Participants) | 6 | 4 | 4 | 6
  Percent change at Day 2 | 278.1 (163.60) | 461.6 (175.95) | 708.5 (200.76) | -9.8 (31.29)
  Percent change at Day 7: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 7 | 129.8 (71.07) | 164.3 (114.69) | 306.5 (45.29) | 19.6 (58.46)
  Percent change at Day 14: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 14 | 59.7 (38.36) | 121.1 (132.70) | 163.7 (37.92) | 21.2 (47.33)
  Percent change at Day 19: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 19 | 43.0 (20.81) | 87.2 (92.62) | 153.3 (25.60) | 20.9 (49.01)
  Percent change at Day 28: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 28 | 15.9 (14.37) | 36.5 (57.79) | 157.6 (103.15) | -2.6 (18.74)
  Percent change at Day 45: number analyzed (Participants) | 6 | 5 | 5 | 6
  Percent change at Day 45 | 92.5 (17.60) | 118.9 (116.56) | 267.5 (59.75) | -7.7 (30.53)
  Percent change at Day 56: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 56 | 55.8 (34.06) | 102.2 (74.51) | 220.4 (62.44) | -10.7 (36.98)
  Percent change at Day 75: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 75 | 87.8 (38.89) | 172.1 (141.94) | 314.3 (75.17) | -23.6 (27.01)
  Percent change at Day 84: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 84 | 77.0 (16.80) | 146.3 (146.97) | 224.2 (40.97) | -12.4 (34.64)
  Percent change at Day 103: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 103 | 128.9 (42.92) | 207.3 (159.23) | 315.3 (127.45) | -16.7 (29.36)
  Percent change at Day 112: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 112 | 83.2 (46.16) | 207.4 (176.39) | 275.2 (92.55) | -20.2 (21.83)
  Percent change at Day 131: number analyzed (Participants) | 6 | 6 | 4 | 5
  Percent change at Day 131 | 168.4 (41.44) | 249.0 (204.05) | 393.6 (66.08) | -21.1 (25.48)
  Percent change at Pre-dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Pre-dose Day 140 | 111.1 (25.89) | 185.8 (164.10) | 297.3 (48.94) | 0.2 (68.99)
  Percent change at 1 H Post dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at 1 H Post dose Day 140 | 264.4 (55.03) | 345.7 (201.63) | 553.7 (122.06) | -24.0 (24.14)
  Percent change at 2 H Post dose Day 140: number analyzed (Participants) | 6 | 6 | 4 | 4
  Percent change at 2 H Post dose Day 140 | 337.7 (67.82) | 394.6 (196.64) | 637.8 (146.28) | -28.8 (33.79)
  Percent change at 4 H Post dose Day 140: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at 4 H Post dose Day 140 | 397.0 (70.71) | 459.8 (234.24) | 781.5 (165.36) | -4.9 (53.65)
  Percent change at Day 141: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 141 | 360.6 (70.15) | 539.2 (291.07) | 889.4 (267.61) | -31.3 (20.95)
  Percent change at Day 154: number analyzed (Participants) | 0 | 6 | 5 | 4
  Percent change at Day 154 |  | 241.5 (196.56) | 506.2 (142.03) | -32.3 (22.75)
  Percent change at Day 168: number analyzed (Participants) | 6 | 6 | 5 | 5
  Percent change at Day 168 | 119.7 (30.44) | 176.4 (159.42) | 366.6 (91.33) | -22.8 (27.34)
  Percent change at Day 224: number analyzed (Participants) | 6 | 6 | 5 | 6
  Percent change at Day 224 | 29.7 (37.85) | 27.1 (74.59) | 102.6 (41.52) | 8.2 (68.87)
  Percent change at Day 304 / ET: number analyzed (Participants) | 0 | 6 | 5 | 3
  Percent change at Day 304 / ET |  | 15.4 (66.96) | 11.0 (12.78) | -38.8 (22.12)

23. Secondary Outcome: Change From Baseline in Vital Signs at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET: Systolic and Diastolic Blood Pressure
Time Frame: Baseline, 1 and 4 hour (H) post-dose on Day 1; 24 H post-dose on Days 2 and 141; pre-dose and 4 - 8 H post-dose on Days 28, 56, 84, 112; pre-dose and 1, 4 H post-dose on Day 140; Day 7, 14, 19, 45, 75, 103;131, 141, 154 168, 224 and 304/ET
Population: Safety analysis set included all randomized participants who received any amount of study drug. Here "Number Analyzed" signifies number of participants evaluated for given time point.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
millimeter of mercury (mmHg)
  Baseline: SBP | 128.0 (10.58) | 128.7 (18.05) | 127.3 (7.37) | 125.3 (12.19)
  Change at 1H post-dose Day 1: SBP | 11.3 (10.71) | -5.7 (16.56) | 3.8 (11.70) | 2.5 (6.38)
  Change at 4 H post-dose Day 1: SBP | 1.0 (8.56) | -1.3 (17.42) | 2.2 (9.64) | 2.7 (12.55)
  Change at 24 H post-dose Day 2: SBP | 5.0 (11.22) | -10.7 (18.53) | -5.0 (8.29) | 0.8 (4.62)
  Change at Day 7: SBP | 7.3 (22.08) | -5.3 (15.47) | -1.5 (7.74) | -4.0 (4.15)
  Change at Day 14: SBP | 2.0 (15.13) | -1.5 (9.29) | -7.2 (11.84) | 2.8 (7.49)
  Change at Day 19: SBP: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 19: SBP | -1.3 (7.45) | -6.2 (9.43) | -8.6 (8.35) | -1.3 (3.20)
  Change at pre-dose Day 28: SBP | 7.7 (11.83) | -8.8 (10.09) | -1.3 (11.76) | -0.3 (9.56)
  Change at 4-8 H post-dose Day 28: SBP: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at 4-8 H post-dose Day 28: SBP | 7.7 (10.61) | -5.5 (12.29) | 3.6 (11.80) | 7.3 (18.69)
  Change at Day 45: SBP: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 45: SBP | 3.7 (6.62) | 0.3 (12.31) | -1.6 (23.42) | 4.3 (7.12)
  Change at pre-dose Day 56: SBP | 5.0 (15.48) | -1.3 (9.61) | -4.5 (14.71) | 3.2 (9.52)
  Change at 4-8 H post-dose day 56: SBP: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 4-8 H post-dose day 56: SBP | 4.8 (10.82) | -1.7 (7.34) | -0.2 (11.58) | 8.2 (17.48)
  Change at Day 75: SBP: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 75: SBP | -0.7 (19.34) | -1.8 (16.57) | 1.8 (15.88) | 6.0 (11.77)
  Change at Pre-dose Day 84: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Pre-dose Day 84: SBP | 3.2 (15.05) | -0.8 (8.91) | -0.3 (15.88) | 10.0 (9.67)
  Change at 4-8H post-dose Day 84: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4-8H post-dose Day 84: SBP | 0.0 (9.63) | -7.0 (12.62) | 3.8 (10.30) | 7.0 (13.58)
  Change at Day 103: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 103: SBP | 2.0 (13.08) | -1.3 (11.29) | 5.5 (8.62) | 11.4 (12.03)
  Change at pre-dose Day 112: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112: SBP | -2.0 (12.65) | -1.2 (17.28) | -0.5 (10.35) | 12.8 (8.87)
  Change at 4-8 H post-dose Day 112: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4-8 H post-dose Day 112: SBP | -4.7 (8.26) | -2.7 (10.25) | -1.7 (11.64) | 7.4 (14.62)
  Change at Day 131: SBP: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 131: SBP | 4.3 (13.11) | 0.2 (12.59) | 1.0 (9.75) | 12.2 (13.20)
  Change at pre-dose Day 140: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140: SBP | -5.3 (15.78) | -2.3 (16.42) | -2.8 (8.16) | 2.6 (8.56)
  Change at 1 H post-dose Day 140: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140: SBP | -0.7 (11.64) | -1.3 (12.75) | -1.0 (13.71) | 5.4 (20.51)
  Change at 4 H post dose Day 140: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140: SBP | -6.0 (9.96) | -6.7 (16.44) | -3.3 (8.57) | 12.4 (7.44)
  Change at 24 H post dose Day 141: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 24 H post dose Day 141: SBP | -6.0 (11.10) | -2.5 (10.43) | -0.7 (3.33) | 10.2 (11.99)
  Change at Day 154: SBP: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 154: SBP |  | -2.7 (8.80) | -6.7 (8.24) | 0.3 (7.41)
  Change at Day 168: SBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: SBP | 5.8 (24.04) | -0.8 (11.18) | -11.8 (7.96) | 5.2 (11.12)
  Change at Day 224/ET: SBP | 1.8 (15.83) | 4.7 (14.88) | -3.0 (12.81) | 5.5 (9.93)
  Change at Day 304/ET: SBP: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: SBP |  | -1.7 (9.07) | 0.5 (18.57) | 2.3 (15.52)
  Baseline: DBP | 78.7 (7.55) | 75.0 (10.56) | 80.3 (7.74) | 76.7 (5.99)
  Change at 1 H post-dose Day 1: DBP | -0.3 (7.09) | 3.5 (9.38) | 3.0 (8.44) | -3.3 (7.26)
  Change at 4 H post-dose Day 1: DBP | -3.7 (11.48) | -1.5 (8.09) | 0.2 (8.01) | -4.3 (4.03)
  Change at 24 H post-dose Day 2: DBP | -2.7 (8.36) | -0.7 (5.32) | -4.7 (8.80) | -2.2 (8.82)
  Change at Day 7: DBP | -1.7 (11.48) | 4.7 (8.26) | -2.7 (9.44) | -2.3 (6.47)
  Change at Day 14: DBP | -1.3 (6.02) | 3.7 (9.91) | -3.7 (10.63) | -1.3 (6.06)
  Change at Day 19: DBP: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 19: DBP | -1.7 (7.84) | -1.2 (6.59) | -5.4 (4.45) | -3.7 (6.83)
  Change at pre-dose Day 28: DBP | -1.0 (11.51) | -2.2 (8.95) | -2.8 (11.72) | -4.8 (8.16)
  Change at 4-8 H post-dose Day 28:DBP: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at 4-8 H post-dose Day 28:DBP | 0.7 (6.53) | 0.0 (12.90) | 2.6 (4.22) | -4.5 (7.15)
  Change at Day 45: DBP: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 45: DBP | 1.7 (5.99) | 5.8 (11.74) | -4.6 (11.99) | -2.0 (10.97)
  Change at pre-dose Day 56: DBP | 1.0 (5.33) | 0.3 (10.98) | -1.0 (5.06) | 2.3 (8.73)
  Change at 4-8 H post-dose day 56: DBP: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 4-8 H post-dose day 56: DBP | 0.8 (5.00) | -0.5 (11.93) | 1.4 (7.20) | -3.0 (6.44)
  Change at Day 75: DBP: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 75: DBP | -0.3 (6.12) | -3.2 (10.01) | -4.6 (5.59) | -1.2 (6.53)
  Change at pre-dose Day 84: DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 84: DBP | -0.7 (8.45) | 0.8 (14.76) | -1.2 (11.39) | 2.2 (7.66)
  Change at 4-8 H post-dose Day 84:DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4-8 H post-dose Day 84:DBP | -6.7 (7.97) | -3.0 (8.07) | 0.5 (10.25) | -2.0 (6.67)
  Change at Day 103: DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 103: DBP | -5.0 (5.76) | 0.3 (12.23) | 2.2 (7.96) | 3.4 (4.04)
  Change at pre-dose Day 112: DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112: DBP | -1.8 (8.35) | 3.3 (10.80) | -2.3 (5.01) | 4.4 (4.39)
  Change at 4-8 H post-dose Day 112:DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4-8 H post-dose Day 112:DBP | -1.3 (8.16) | 0.0 (10.73) | -1.0 (6.93) | 1.0 (7.55)
  Change at Day 131: DBP: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 131: DBP | -1.3 (3.01) | -1.7 (8.48) | -3.4 (8.99) | 0.0 (5.34)
  Change at pre-dose Day 140: DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140: DBP | -4.3 (10.15) | 2.5 (11.20) | 1.0 (14.52) | -0.4 (5.32)
  Change at 1 H post-dose Day 140: DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140: DBP | -2.7 (7.87) | 4.2 (10.82) | -1.3 (10.19) | -2.2 (6.22)
  Change at 4 H post dose Day 140: DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140: DBP | -6.3 (8.24) | 3.3 (9.20) | -6.5 (8.24) | -2.2 (5.22)
  Change at 24 H post dose Day 141: DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 24 H post dose Day 141: DBP | -4.7 (4.13) | 2.2 (12.04) | -4.5 (7.09) | 0.6 (6.73)
  Change at Day 154: DBP: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 154: DBP |  | 2.5 (8.85) | -5.5 (5.79) | -4.0 (4.97)
  Change at Day 168: DBP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: DBP | -2.2 (6.88) | 0.0 (11.51) | -4.8 (7.00) | 1.0 (5.92)
  Change at Day 224/ET: DBP | -0.8 (8.50) | 1.0 (8.00) | -3.0 (4.52) | -0.5 (5.96)
  Change at Day 304/ET: DBP: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: DBP |  | 1.3 (11.57) | 1.2 (16.41) | 2.8 (4.99)

24. Secondary Outcome: Change From Baseline in Vital Signs at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET: Pulse Rate
Time Frame: Baseline, 1 and 4 H post-dose on Day 1; 24 H post-dose on Days 2 and 141; pre-dose and 4 - 8 H post-dose on Days 28, 56, 84, 112; pre-dose and 1, 4 H post-dose on Day 140; Day 7, 14, 19, 45, 75, 103;131, 141, 154 168, 224 and 304/ET
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Beats per minute
  Baseline | 64.2 (6.40) | 62.8 (4.40) | 66.5 (6.53) | 66.7 (5.01)
  Change at 1H post-dose Day 1 | 1.7 (2.66) | -1.8 (4.40) | -4.2 (5.46) | 1.0 (8.83)
  Change at 4 H post-dose Day 1 | 3.5 (6.25) | 1.2 (5.81) | -2.3 (7.50) | 4.0 (7.77)
  Change at 24 H post-dose Day 2 | 0.8 (2.71) | 1.5 (1.97) | -2.0 (3.74) | 3.8 (6.40)
  Change at Day 7 | 4.5 (3.67) | 3.3 (3.08) | -4.2 (5.42) | 4.2 (5.95)
  Change at Day 14 | 1.2 (2.04) | 4.3 (7.39) | 0.3 (4.59) | 6.0 (6.93)
  Change at Day 19: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 19 | 2.5 (5.92) | 7.8 (7.60) | 0.0 (2.45) | 1.0 (5.76)
  Change at pre-dose Day 28 | 0.2 (5.53) | 2.3 (5.32) | -1.5 (5.72) | -1.2 (2.71)
  Change at 4-8 H post-dose Day 28: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at 4-8 H post-dose Day 28 | 6.5 (10.15) | 2.2 (2.56) | -2.8 (4.32) | 0.3 (12.04)
  Change at Day 45: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 45 | 3.5 (2.17) | 2.3 (4.03) | 5.2 (7.26) | -3.0 (5.73)
  Change at pre-dose Day 56 | 1.2 (2.99) | 1.5 (4.37) | -3.7 (5.13) | 2.0 (5.51)
  Change at 4-8 H post-dose day 56: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 4-8 H post-dose day 56 | 3.0 (4.69) | 2.3 (4.13) | 1.6 (10.14) | 6.0 (9.08)
  Change at Day 75: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 75 | 1.5 (4.64) | 5.5 (6.19) | 8.0 (8.12) | 6.8 (8.90)
  Change at pre-dose Day 84: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 84 | 2.3 (3.83) | 4.0 (3.10) | -1.8 (4.17) | 2.2 (7.09)
  Change at 4-8 H post-dose Day 84: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4-8 H post-dose Day 84 | -0.3 (5.89) | 1.8 (4.31) | -2.7 (7.76) | 4.2 (5.12)
  Change at Day 103: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 103 | 2.2 (2.04) | 2.5 (4.09) | 1.3 (1.63) | 6.0 (5.29)
  Change at pre-dose Day 112: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112 | -0.8 (4.02) | 1.5 (3.33) | -0.2 (4.26) | 0.2 (5.02)
  Change at 4-8 H post-dose Day 112: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4-8 H post-dose Day 112 | 1.8 (2.86) | 3.3 (5.05) | -2.2 (3.19) | -1.6 (0.89)
  Change at Day 131: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 131 | 1.8 (4.07) | 7.2 (7.55) | 2.8 (13.07) | 1.8 (6.94)
  Change at pre-dose Day 140: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140 | 2.5 (3.99) | 2.8 (4.07) | -0.8 (4.79) | 3.2 (3.27)
  Change at 1 H post-dose Day 140: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140 | -0.5 (4.37) | 0.8 (5.53) | -4.5 (6.83) | -3.2 (9.09)
  Change at 4 H post dose Day 140.: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140. | 3.2 (4.83) | 4.0 (8.94) | -2.8 (6.91) | -1.0 (10.20)
  Change at 24 H post dose Day 141: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 24 H post dose Day 141 | 1.0 (3.22) | 8.7 (3.88) | -2.0 (6.10) | 6.4 (4.77)
  Change at Day 154: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 154 |  | 9.2 (3.82) | 0.5 (8.73) | 13.5 (5.00)
  Change at Day 168: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168 | 1.7 (1.86) | -0.5 (4.89) | -6.8 (5.42) | 4.8 (7.56)
  Change at Day 224/ET | -1.2 (6.94) | 0.3 (5.01) | -0.7 (5.99) | 0.5 (4.55)
  Change at Day 304/ET: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET |  | 1.2 (5.88) | -0.2 (2.56) | 2.0 (5.66)

25. Secondary Outcome: Change From Baseline in Vital Signs at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET: Temperature
Time Frame: as for outcome 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Degree Celsius
  Baseline | 36.40 (0.228) | 36.72 (0.256) | 36.87 (0.082) | 36.72 (0.397)
  Change at 1H post-dose Day 1 | 0.30 (0.405) | 0.10 (0.253) | -0.10 (0.190) | 0.08 (0.183)
  Change at 4 H post-dose Day 1 | 0.18 (0.571) | 0.08 (0.133) | 0.03 (0.207) | 0.17 (0.327)
  Change at 24 H post-dose Day 2 | 0.22 (0.204) | 0.12 (0.232) | -0.32 (0.371) | -0.08 (0.515)
  Change at Day 7 | 0.15 (0.226) | 0.05 (0.315) | -0.40 (0.405) | 0.00 (0.276)
  Change at Day 14 | 0.37 (0.350) | -0.03 (0.327) | 0.08 (0.117) | 0.05 (0.243)
  Change at Day 19: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 19 | 0.43 (0.234) | -0.12 (0.271) | 0.04 (0.288) | -0.02 (0.183)
  Change at pre-dose Day 28 | 0.18 (0.204) | -0.10 (0.283) | -0.02 (0.172) | -0.17 (0.294)
  Change at 4-8 H post-dose Day 28: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at 4-8 H post-dose Day 28 | 0.28 (0.172) | 0.15 (0.339) | 0.00 (0.158) | 0.03 (0.186)
  Change at Day 45: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 45 | 0.13 (0.413) | 0.12 (0.483) | -0.06 (0.195) | 0.03 (0.516)
  Change at pre-dose Day 56 | 0.05 (0.476) | 0.08 (0.366) | 0.03 (0.175) | 0.07 (0.350)
  Change at 4-8 H post-dose day 56: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at 4-8 H post-dose day 56 | 0.22 (0.313) | 0.13 (0.273) | 0.12 (0.084) | 0.00 (0.436)
  Change at Day 75: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 75 | -0.15 (0.437) | 0.07 (0.333) | -0.06 (0.279) | -0.28 (0.383)
  Change at pre-dose Day 84: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 84 | -0.03 (0.216) | -0.03 (0.320) | 0.02 (0.147) | -0.10 (0.400)
  Change at 4-8 H post-dose Day 84: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4-8 H post-dose Day 84 | -0.13 (0.665) | 0.00 (0.167) | 0.03 (0.103) | 0.10 (0.274)
  Change at Day 103: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 103 | 0.05 (0.394) | -0.08 (0.462) | -0.10 (0.219) | -0.06 (0.251)
  Change at pre-dose Day 112: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112 | -0.08 (0.512) | 0.12 (0.279) | -0.15 (0.274) | -0.20 (0.292)
  Change at 4-8 H post-dose Day 112: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4-8 H post-dose Day 112 | 0.03 (0.437) | 0.12 (0.387) | -0.22 (0.293) | 0.06 (0.336)
  Change at Day 131: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 131 | 0.18 (0.387) | 0.02 (0.458) | -0.14 (0.288) | -0.04 (0.261)
  Change at pre-dose Day 140: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140 | 0.10 (0.352) | -0.05 (0.432) | -0.07 (0.207) | -0.02 (0.311)
  Change at 1 H post-dose Day 140: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140 | 0.02 (0.496) | 0.08 (0.407) | -0.03 (0.197) | -0.30 (0.224)
  Change at 4 H post dose Day 140: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140 | 0.23 (0.197) | 0.05 (0.428) | -0.12 (0.248) | -0.14 (0.270)
  Change at 24 H post dose Day 141: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 24 H post dose Day 141 | 0.00 (0.210) | 0.08 (0.248) | -0.18 (0.183) | -0.14 (0.365)
  Change at Day 154: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 154 |  | 0.07 (0.266) | -0.25 (0.414) | 0.00 (0.141)
  Change at Day 168: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168 | 0.27 (0.459) | -0.12 (0.293) | -0.18 (0.264) | 0.12 (0.192)
  Change at Day 224/ET | 0.03 (0.446) | 0.07 (0.234) | -0.07 (0.288) | 0.03 (0.472)
  Change at Day 304/ET: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET |  | -0.10 (0.283) | -0.10 (0.167) | -0.08 (0.150)

26. Secondary Outcome: Change From Baseline in Vital Signs at Day 1, 2, 7, 14, 19, 28, 45, 56, 75, 84, 103, 112, 131, 140, 141, 154, 168, 224, 304/ET: Weight
Time Frame: as for outcome 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Kilogram
  Baseline | 81.74 (9.975) | 85.85 (8.443) | 78.58 (12.497) | 80.14 (21.430)
  Change at Day 19: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 19 | 0.25 (0.709) | -0.05 (1.588) | 0.09 (1.330) | 0.93 (0.945)
  Change at Day 28 | 0.46 (0.749) | -0.12 (2.098) | 0.02 (1.172) | 0.29 (0.661)
  Change at Day 45: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 45 | 0.71 (1.654) | -0.49 (2.298) | 0.52 (0.899) | 0.36 (1.219)
  Change at Day 56 | 0.72 (1.425) | -0.99 (2.371) | -1.21 (2.942) | 0.52 (0.616)
  Change at Day 75: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 75 | 0.60 (1.464) | -0.46 (3.267) | 0.48 (0.883) | 0.98 (0.641)
  Change at Day 84: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84 | 0.63 (1.538) | -0.54 (3.194) | -0.16 (0.943) | 0.99 (1.050)
  Change at Day 103: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 103 | -0.60 (4.787) | -0.75 (3.213) | 0.22 (1.249) | 1.23 (1.490)
  Change at Day 112: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112 | 0.67 (1.118) | 0.05 (3.638) | -0.05 (0.731) | 1.43 (1.097)
  Change at Day 131: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 131 | 1.35 (1.354) | -0.43 (4.197) | -0.08 (0.646) | 1.67 (1.159)
  Change at Day 140: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140 | 1.06 (0.833) | -0.36 (4.233) | -0.46 (1.248) | 1.37 (1.708)
  Change at Day 154: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 154 |  | -3.78 (8.246) | -0.57 (1.301) | 1.03 (1.464)
  Change at Day 168: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168 | 1.74 (2.723) | -1.35 (4.393) | -0.84 (1.237) | 1.26 (1.312)
  Change at Day 224/ ET | 0.85 (0.976) | -1.97 (4.284) | 1.49 (4.376) | 1.42 (1.679)
  Change at Day 304/ET: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET |  | 0.71 (6.545) | 3.04 (4.327) | 0.60 (0.678)

27. Secondary Outcome: Change From Baseline Electrocardiogram (ECG) 12-lead at Day 1, 28, 56, 84, 112, 140, 168, 224, 304/ET
Description: Criteria for changes in ECG (12-lead) were defined as: PR interval >=220 millisecond (msec) and increase of >=20 msec; QRS interval >=120 msec; QT interval corrected using the Bazett's formula (QTcB) >=500 msec; Maximum Change from Baseline in QTcF at Borderline >=30 msec to <60 msec and Prolonged >=60 msec.
Time Frame: Baseline, 1 and 4 H post-dose on Day 1; pre-dose on Days 28, 56, 84, 112; pre-dose and 1, 4 H post-dose on Day 140; Day 168, 224 and 304/ET
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Millisecond
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Millisecond
  Baseline: RR | 939.28 (124.486) | 962.44 (117.246) | 918.39 (101.325) | 928.33 (117.701)
  Change at 1 H post-dose Day 1: RR | 4.06 (45.449) | 24.94 (70.632) | 79.11 (89.729) | -21.22 (136.555)
  Change at 4 H post-dose Day 1: RR | -36.28 (38.148) | -34.22 (82.327) | 22.33 (115.576) | -54.11 (94.978)
  Change at pre-dose Day 28: RR | 29.56 (40.059) | 0.39 (53.575) | 69.44 (91.732) | 49.00 (78.316)
  Change at pre-dose Day 56: RR | 5.39 (61.533) | -19.78 (32.654) | 74.78 (98.804) | 8.83 (65.440)
  Change at pre-dose Day 84: RR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 84: RR | -7.61 (53.735) | -12.78 (56.646) | 57.11 (102.514) | -51.67 (186.668)
  Change at pre-dose Day 112: RR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112: RR | 30.56 (23.478) | -24.11 (63.637) | 34.94 (77.744) | -44.87 (82.091)
  Change at pre-dose Day 140: RR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140: RR | -6.39 (43.272) | -39.89 (85.486) | 26.56 (91.107) | -9.60 (51.462)
  Change at 1 H post-dose Day 140: RR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140: RR | -6.78 (120.518) | -16.83 (58.974) | 80.44 (104.487) | 42.60 (150.052)
  Change at 4 H post dose Day 140: RR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140: RR | -44.61 (76.284) | -66.17 (86.676) | 52.17 (86.145) | 5.13 (166.054)
  Change at Day 168: RR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: RR | -33.11 (80.934) | -31.78 (27.507) | 60.44 (122.291) | -28.67 (70.982)
  Change at Day 224/ET: RR | 21.72 (77.289) | 8.89 (58.224) | -22.72 (99.733) | 56.50 (78.870)
  Change at Day 304/ET: RR: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: RR |  | 32.39 (70.600) | -9.22 (80.263) | -11.92 (122.446)
  Baseline: PR | 170.78 (23.268) | 190.00 (38.006) | 167.89 (25.711) | 166.11 (41.177)
  Change at 1 H post-dose Day 1: PR | -4.22 (13.589) | -4.33 (9.407) | -7.11 (12.261) | -2.67 (6.902)
  Change at 4 H post-dose Day 1: PR | -1.33 (9.762) | -4.89 (6.898) | -6.33 (7.563) | -2.89 (6.362)
  Change at pre-dose Day 28: PR | -2.78 (11.711) | 1.00 (10.673) | 28.44 (84.486) | 3.89 (12.245)
  Change at pre-dose Day 56: PR: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at pre-dose Day 56: PR | -6.78 (9.270) | 0.33 (15.842) | -11.47 (22.912) | 12.22 (23.512)
  Change at pre-dose Day 84: PR: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at pre-dose Day 84: PR | 0.22 (6.885) | -8.33 (18.426) | -0.67 (1.944) | 11.73 (32.392)
  Change at pre-dose Day 112: PR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112: PR | -0.78 (12.567) | -3.33 (18.086) | -13.56 (22.134) | 16.53 (26.764)
  Change at pre-dose Day 140: PR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140: PR | 2.33 (8.892) | -1.11 (14.052) | -4.22 (5.311) | 11.33 (23.636)
  Change at 1 H post-dose Day 140: PR: number analyzed (Participants) | 5 | 6 | 6 | 5
  Change at 1 H post-dose Day 140: PR | -3.33 (7.760) | -1.56 (11.938) | -4.67 (14.569) | 16.27 (22.229)
  Change at 4 H post dose Day 140: PR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140: PR | -4.33 (9.177) | 2.00 (8.316) | -7.89 (11.262) | 21.87 (28.757)
  Change at Day 168: PR: number analyzed (Participants) | 6 | 6 | 6 | 4
  Change at Day 168: PR | -4.11 (8.405) | -7.00 (12.994) | -2.56 (5.154) | -1.50 (10.932)
  Change at Day 224/ET: PR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: PR | -7.11 (14.090) | -1.00 (15.468) | -7.89 (7.061) | 14.13 (24.214)
  Change at Day 304/ET: PR: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: PR |  | -3.00 (19.066) | -17.22 (21.935) | 16.33 (21.709)
  Baseline: QRS | 87.11 (5.036) | 91.44 (8.352) | 97.89 (22.444) | 100.33 (24.858)
  Change at 1 H post-dose Day 1: QRS | -2.67 (4.881) | -1.56 (3.417) | -2.33 (2.789) | 0.78 (1.760)
  Change at 4 H post-dose Day 1: QRS | -1.78 (4.856) | -1.67 (2.692) | 0.44 (2.373) | 0.78 (3.410)
  Change at pre-dose Day 28: QRS | 1.56 (4.375) | -1.44 (3.410) | -0.89 (2.656) | -0.33 (2.261)
  Change at pre-dose Day 56: QRS | -1.44 (2.083) | 0.22 (5.054) | 1.78 (2.722) | -2.67 (6.037)
  Change at pre-dose Day 84: QRS: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 84: QRS | -2.11 (3.331) | -0.11 (6.217) | 6.78 (22.333) | 1.60 (9.541)
  Change at pre-dose Day 112: QRS: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112: QRS | -3.11 (7.101) | 1.56 (4.593) | 5.11 (20.149) | 0.80 (4.840)
  Change at pre-dose Day 140: QRS: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140: QRS | -2.67 (4.638) | 1.22 (5.439) | 0.33 (2.883) | -0.40 (4.017)
  Change at 1 H post-dose Day 140: QRS: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140: QRS | -2.56 (3.538) | 0.67 (6.613) | 1.22 (2.083) | 0.40 (4.681)
  Change at 4 H post dose Day 140: QRS: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140: QRS | -2.22 (3.202) | -0.22 (4.456) | -0.44 (1.440) | 2.53 (5.586)
  Change at Day 168: QRS: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: QRS | -4.44 (5.106) | 1.89 (5.340) | 2.11 (4.530) | 0.00 (4.922)
  Change at Day 224/ET: QRS | -2.44 (6.017) | 0.22 (3.569) | 9.78 (26.712) | 1.00 (2.692)
  Change at Day 304/ET: QRS: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: QRS |  | 1.22 (6.895) | -2.56 (1.760) | 5.83 (4.631)
  Baseline: QT | 405.00 (25.174) | 422.00 (29.835) | 408.56 (30.560) | 401.78 (31.932)
  Change at 1H post-dose Day 1: QT | 1.22 (14.270) | 2.22 (11.713) | 14.22 (14.845) | 0.78 (26.346)
  Change at 4 H post-dose Day 1: QT | -3.78 (18.493) | -13.44 (19.018) | 4.67 (29.796) | 1.56 (32.457)
  Change at pre-dose Day 28: QT | -1.33 (13.367) | -11.33 (17.420) | 11.11 (14.228) | 4.89 (18.290)
  Change at pre-dose Day 56: QT | -2.33 (11.939) | -8.67 (10.302) | 18.44 (31.865) | 8.22 (10.221)
  Change at pre-dose Day 84: QT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 84: QT | -2.33 (15.769) | -11.33 (13.914) | 14.11 (26.319) | 10.27 (28.482)
  Change at pre-dose Day 112: QT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112: QT | -1.00 (5.379) | -9.33 (17.420) | 5.44 (13.607) | 19.07 (35.345)
  Change at pre-dose Day 140: QT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140: QT | -3.44 (12.274) | -6.00 (14.092) | 11.89 (18.621) | 7.47 (25.304)
  Change at 1 H post-dose Day 140: QT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140: QT | -4.67 (24.909) | -18.00 (35.700) | 22.33 (22.170) | 19.33 (28.091)
  Change at 4 H post dose Day 140: QT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140: QT | -10.22 (12.174) | -13.00 (17.006) | 19.67 (14.340) | 11.33 (35.308)
  Change at Day 168: QT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: QT | -13.00 (17.255) | -5.67 (11.939) | 16.44 (36.302) | 4.27 (26.594)
  Change at Day 224/ET: QT | -1.67 (6.782) | -9.67 (12.442) | -1.22 (27.995) | 19.22 (22.225)
  Change at Day 304/ET: QT: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: QT |  | -1.67 (16.896) | -8.56 (31.792) | 9.33 (36.127)
  Baseline: QTcB | 418.56 (13.605) | 430.67 (20.976) | 426.28 (18.370) | 417.11 (17.539)
  Change at 1 H post-dose Day 1: QTcB | 0.39 (4.823) | -3.50 (6.483) | -2.67 (12.006) | 5.81 (17.269)
  Change at 4 H post-dose Day 1: QTcB | 4.44 (13.274) | -6.67 (14.188) | -0.11 (6.811) | 13.50 (29.257)
  Change at pre-dose Day 28: QTcB | -6.39 (17.989) | -12.50 (14.442) | -2.94 (18.639) | -5.94 (5.953)
  Change at pre-dose Day 56: QTcB | -2.06 (16.679) | -4.67 (9.920) | 1.56 (15.450) | 5.39 (19.841)
  Change at pre-dose Day 84: QTcB: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 84: QTcB | -0.89 (8.516) | -9.33 (16.350) | 2.22 (21.281) | 23.07 (32.116)
  Change at pre-dose Day 112: QTcB: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112: QTcB | -6.89 (9.135) | -4.33 (8.899) | -1.11 (9.660) | 29.07 (42.361)
  Change at pre-dose Day 140: QTcB: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140: QTcB | -2.11 (6.493) | 3.17 (11.201) | 6.94 (6.641) | 9.33 (22.955)
  Change at 1 H post-dose Day 140: QTcB: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140: QTcB | -0.61 (9.855) | -14.78 (38.322) | 4.72 (10.794) | 11.33 (18.318)
  Change at 4 H post dose Day 140: QTcB: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140: QTcB | 0.72 (9.525) | 1.83 (9.697) | 9.06 (11.144) | 11.80 (20.895)
  Change at Day 168: QTcB: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: QTcB | -6.39 (18.637) | 1.33 (13.471) | 4.06 (10.810) | 10.07 (21.177)
  Change at Day 224/ET: QTcB | -5.39 (11.496) | -12.33 (13.105) | 3.72 (14.188) | 6.72 (17.425)
  Change at Day 304/ET: QTcB: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: QTcB |  | -9.5 (15.812) | -6.28 (17.655) | 13.17 (8.813)

28. Secondary Outcome: Change From Baseline in Heart Rate at Day 1, 28, 56, 84, 112, 140, 168, 224, 304/ET
Time Frame: as for outcome 27
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Beats per minute
  Baseline | 64.94 (9.318) | 63.17 (7.327) | 66.06 (7.295) | 65.44 (7.556)
  Change at 1 H post-dose Day 1 | -0.33 (3.026) | -1.67 (4.142) | -5.44 (6.527) | 2.72 (10.603)
  Change at 4 H post-dose Day 1 | 2.28 (2.752) | 2.11 (5.188) | -1.72 (8.045) | 4.00 (7.226)
  Change at pre-dose Day 28 | -1.78 (2.562) | -0.17 (3.475) | -4.39 (5.463) | -3.78 (5.496)
  Change at pre-dose Day 56 | 0.39 (4.096) | 1.17 (1.810) | -4.89 (7.290) | -1.11 (4.617)
  Change at pre-dose Day 84: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 84 | 0.22 (3.410) | 0.50 (3.378) | -3.72 (6.191) | 4.00 (12.243)
  Change at pre-dose Day 112: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112 | -1.78 (1.559) | 1.33 (4.580) | -1.89 (3.959) | 3.00 (6.342)
  Change at pre-dose Day 140: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140 | 0.50 (2.606) | 2.89 (5.556) | -1.39 (6.591) | 0.93 (3.919)
  Change at 1 H post-dose Day 140: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140 | 2.61 (11.432) | 1.17 (3.650) | -5.22 (6.649) | -2.13 (10.038)
  Change at 4 H post dose Day 140: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140 | 3.67 (5.578) | 5.11 (6.869) | -3.61 (5.752) | 0.47 (12.613)
  Change at Day 168: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168 | 2.22 (5.419) | 2.00 (1.687) | -3.56 (7.745) | 2.20 (5.316)
  Change at Day 224/ET | -0.61 (5.031) | -0.67 (4.279) | 1.11 (7.067) | -3.44 (5.730)
  Change at Day 304/ET: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET |  | -2.50 (4.451) | 0.94 (6.220) | 3.08 (9.094)

29. Secondary Outcome: Change From Baseline in Bilirubin, Direct Bilirubin, Blood Urea Nitrogen, Creatinine, Uric Acid, Calcium, Phosphate, Glucose, Cholesterol, Triglycerides, Immunoglobulin G, Immunoglobulin A, Immunoglobulin M at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Description: Following parameters were analyzed for laboratory examination: Bilirubin, Direct Bilirubin, Blood Urea Nitrogen(BUN), Creatinine, Uric Acid, Calcium, Phosphate, Glucose, Cholesterol (CL)(Fasting), Triglycerides (Fasting) (TG), Immunoglobulin G (Ig G), Immunoglobulin A (Ig A), Immunoglobulin M (Ig M)
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: All randomized participants who met the inclusion criteria and received any amount of study drug were included. Here "Number Analyzed" signifies number of participants evaluated for given time point. Categories with at least 1 non-zero data have been provided below.
Measure: Mean (Standard Deviation); unit: Milligram per deciliter (MG/DL)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Milligram per deciliter (MG/DL)
  Baseline: Bilirubin | 0.48 (0.147) | 0.58 (0.422) | 0.47 (0.234) | 0.52 (0.204)
  Change at Day 28: Bilirubin: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Bilirubin | -0.05 (0.122) | -0.12 (0.264) | 0.08 (0.435) | -0.10 (0.126)
  Change at Day 56: Bilirubin | 0.02 (0.133) | -0.07 (0.121) | 0.25 (0.409) | -0.07 (0.121)
  Change at Day 84: Bilirubin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Bilirubin | -0.03 (0.082) | -0.03 (0.250) | 0.12 (0.133) | -0.10 (0.122)
  Change at Day 112: Bilirubin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Bilirubin | -0.10 (0.141) | -0.08 (0.325) | 0.20 (0.276) | -0.10 (0.158)
  Change at Day 140: Bilirubin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Bilirubin | -0.07 (0.082) | -0.02 (0.343) | 0.20 (0.316) | -0.10 (0.158)
  Change at Day 168: Bilirubin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Bilirubin | -0.02 (0.075) | 0.00 (0.200) | 0.17 (0.423) | -0.08 (0.192)
  Change at Day 224/ET: Bilirubin | -0.07 (0.082) | 0.00 (0.210) | 0.02 (0.133) | -0.07 (0.163)
  Change at Day 304/ET: Bilirubin: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Bilirubin |  | 0.05 (0.105) | 0.20 (0.415) | -0.05 (0.100)
  Baseline: Direct Bilirubin | 0.15 (0.055) | 0.17 (0.082) | 0.15 (0.055) | 0.13 (0.052)
  Change at Day 28: Direct Bilirubin: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Direct Bilirubin | -0.03 (0.052) | -0.03 (0.052) | 0.00 (0.082) | -0.02 (0.041)
  Change at Day 56: Direct Bilirubin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 56: Direct Bilirubin | 0.00 (0.063) | 0.00 (0.000) | 0.02 (0.098) | 0.00 (0.071)
  Change at Day 84: Direct Bilirubin: number analyzed (Participants) | 6 | 6 | 6 | 4
  Change at Day 84: Direct Bilirubin | 0.00 (0.063) | -0.02 (0.041) | 0.00 (0.063) | 0.00 (0.000)
  Change at Day 112: Direct Bilirubin: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112: Direct Bilirubin | -0.02 (0.075) | -0.02 (0.041) | 0.00 (0.071) | 0.02 (0.045)
  Change at Day 140: Direct Bilirubin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Direct Bilirubin | -0.03 (0.052) | -0.02 (0.041) | 0.00 (0.063) | 0.00 (0.000)
  Change at Day 168: Direct Bilirubin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Direct Bilirubin | -0.02 (0.041) | -0.02 (0.041) | 0.02 (0.098) | 0.02 (0.045)
  Change at Day 224/ET: Direct Bilirubin | -0.02 (0.075) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.063)
  Change at Day 304/ET: Direct Bilirubin: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Direct Bilirubin |  | 0.00 (0.000) | 0.02 (0.098) | 0.03 (0.050)
  Baseline: BUN | 18.7 (5.01) | 15.5 (3.89) | 18.8 (3.87) | 23.3 (8.33)
  Change at Day 28: BUN: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: BUN | -0.3 (3.14) | -0.2 (2.64) | 0.5 (7.14) | 1.5 (3.73)
  Change at Day 56: BUN | -2.0 (2.10) | -1.2 (4.62) | 2.7 (1.63) | 0.0 (4.52)
  Change at Day 84: BUN: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: BUN | 1.3 (4.32) | 1.3 (3.78) | -0.2 (5.98) | -3.6 (7.02)
  Change at Day 112: BUN: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: BUN | -0.2 (5.08) | -0.5 (2.74) | 1.7 (4.27) | -1.0 (7.62)
  Change at Day 140: BUN: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: BUN | 1.0 (4.60) | -0.2 (4.07) | 1.3 (2.42) | -1.6 (5.41)
  Change at Day 168: BUN: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: BUN | 0.0 (2.45) | 0.5 (3.51) | 1.0 (3.46) | -1.2 (6.76)
  Change at Day 224/ET: BUN | 1.2 (2.14) | 1.3 (2.80) | 0.8 (2.93) | -0.5 (8.87)
  Change at Day 304/ET: BUN: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: BUN |  | 1.5 (2.59) | 2.3 (4.63) | -3.5 (6.35)
  Baseline: Creatinine | 0.918 (0.2322) | 0.955 (0.0750) | 0.917 (0.1657) | 1.105 (0.3136)
  Change at Day 28: Creatinine: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Creatinine | 0.008 (0.1121) | -0.032 (0.0708) | 0.108 (0.1024) | -0.007 (0.1371)
  Change at Day 56: Creatinine | 0.047 (0.0880) | 0.000 (0.1163) | 0.037 (0.0766) | -0.013 (0.1317)
  Change at Day 84: Creatinine: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Creatinine | 0.053 (0.0755) | 0.038 (0.1196) | 0.042 (0.0891) | -0.038 (0.1512)
  Change at Day 112: Creatinine: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Creatinine | 0.043 (0.1179) | 0.008 (0.0924) | 0.082 (0.1389) | -0.024 (0.1747)
  Change at Day 140: Creatinine: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Creatinine | 0.055 (0.1710) | -0.020 (0.1271) | 0.035 (0.0742) | 0.002 (0.1956)
  Change at Day 168: Creatinine: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Creatinine | 0.020 (0.1316) | -0.045 (0.0922) | 0.113 (0.1088) | -0.018 (0.2525)
  Change at Day 224/ET: Creatinine | -0.002 (0.1321) | 0.012 (0.1297) | 0.047 (0.1196) | 0.015 (0.2118)
  Change at Day 304/ET: Creatinine: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Creatinine |  | 0.008 (0.1072) | 0.092 (0.0909) | -0.045 (0.3023)
  Baseline: Uric Acid | 4.87 (1.172) | 5.97 (1.335) | 5.77 (1.039) | 5.58 (1.238)
  Change at Day 28: Uric Acid: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Uric Acid | -0.05 (0.539) | -0.25 (0.176) | 0.03 (0.640) | 0.22 (0.471)
  Change at Day 56: Uric Acid | -0.05 (0.497) | -0.25 (0.383) | 0.00 (0.566) | -0.07 (0.463)
  Change at Day 84: Uric Acid: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Uric Acid | -0.08 (0.722) | 0.07 (0.327) | -0.12 (0.943) | -0.48 (0.487)
  Change at Day 112: Uric Acid: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Uric Acid | -0.32 (0.571) | 0.02 (0.694) | 0.32 (0.804) | 0.10 (0.997)
  Change at Day 140: Uric Acid: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Uric Acid | -0.05 (0.641) | -0.05 (0.701) | 0.18 (0.828) | 0.32 (0.785)
  Change at Day 168: Uric Acid: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Uric Acid | 0.23 (0.855) | -0.03 (0.698) | 0.28 (0.422) | 0.22 (0.779)
  Change at Day 224/ET: Uric Acid | 0.62 (1.072) | 0.07 (0.662) | 0.17 (0.836) | 0.48 (0.933)
  Change at Day 304/ET: Uric Acid: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Uric Acid |  | 0.32 (0.677) | -0.07 (1.143) | -0.10 (0.510)
  Baseline: Calcium | 9.62 (0.248) | 9.62 (0.458) | 9.60 (0.358) | 9.76 (0.301)
  Change at Day 28: Calcium: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Calcium | 0.00 (0.335) | -0.22 (0.264) | -0.02 (0.395) | -0.37 (0.301)
  Change at Day 56: Calcium | 0.17 (0.550) | -0.07 (0.344) | 0.10 (0.540) | -0.22 (0.471)
  Change at Day 84: Calcium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Calcium | 0.10 (0.369) | -0.03 (0.388) | -0.02 (0.387) | -0.38 (0.396)
  Change at Day 112: Calcium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Calcium | -0.17 (0.361) | -0.07 (0.356) | 0.08 (0.488) | -0.26 (0.550)
  Change at Day 140: Calcium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Calcium | 0.13 (0.367) | -0.17 (0.378) | -0.07 (0.472) | -0.16 (0.498)
  Change at Day 168: Calcium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Calcium | -0.15 (0.638) | -0.32 (0.306) | -0.17 (0.327) | -0.30 (0.660)
  Change at Day 224/ET: Calcium | 0.12 (0.279) | -0.27 (0.393) | 0.05 (0.509) | -0.08 (0.512)
  Change at Day 304/ET: Calcium: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Calcium |  | -0.15 (0.446) | 0.23 (0.484) | 0.03 (0.377)
  Baseline: Phosphate | 3.20 (0.583) | 3.48 (0.376) | 3.62 (0.637) | 3.28 (0.717)
  Change at Day 28: Phosphate: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Phosphate | 0.22 (0.417) | 0.08 (0.382) | 0.18 (0.310) | 0.22 (0.508)
  Change at Day 56: Phosphate | -0.03 (0.273) | 0.02 (0.194) | 0.25 (0.539) | 0.22 (0.598)
  Change at Day 84: Phosphate: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Phosphate | 0.27 (0.489) | 0.03 (0.197) | 0.12 (0.512) | 0.12 (0.466)
  Change at Day 112: Phosphate: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Phosphate | 0.27 (0.308) | 0.17 (0.197) | 0.03 (0.356) | 0.38 (0.497)
  Change at Day 140: Phosphate: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Phosphate | 0.32 (0.360) | 0.00 (0.369) | -0.27 (0.575) | 0.58 (0.554)
  Change at Day 168: Phosphate: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Phosphate | 0.17 (0.459) | -0.12 (0.331) | 0.15 (0.418) | 0.36 (0.581)
  Change at Day 224/ET: Phosphate | 0.13 (0.472) | -0.10 (0.456) | 0.15 (0.521) | 0.30 (0.863)
  Change at Day 304/ET: Phosphate: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Phosphate |  | 0.25 (0.217) | 0.12 (0.598) | 0.15 (0.412)
  Baseline: Glucose | 93.8 (11.20) | 92.5 (7.84) | 90.0 (13.97) | 95.8 (9.99)
  Change at Day 28: Glucose: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Glucose | 22.8 (48.16) | 3.8 (9.77) | 7.0 (5.48) | 3.3 (14.39)
  Change at Day 56: Glucose | 1.7 (6.19) | 3.7 (7.42) | 6.5 (15.67) | 0.5 (11.04)
  Change at Day 84: Glucose: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Glucose | -2.0 (1.41) | 7.2 (12.56) | 7.5 (11.47) | 7.8 (13.35)
  Change at Day 112: Glucose: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Glucose | 4.7 (5.28) | 7.3 (12.13) | 9.2 (11.58) | 3.6 (10.67)
  Change at Day 140: Glucose: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Glucose | 6.8 (4.88) | 6.3 (12.04) | 17.7 (7.69) | 11.0 (14.61)
  Change at Day 168: Glucose: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Glucose | -1.0 (6.42) | 3.2 (6.11) | 12.5 (14.79) | 17.6 (32.65)
  Change at Day 224/ET: Glucose | 0.7 (6.28) | 3.3 (5.85) | 8.5 (12.85) | 7.2 (28.03)
  Change at Day 304/ET: Glucose: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Glucose |  | 5.8 (12.16) | 3.8 (15.69) | 20.3 (50.70)
  Baseline: CL (fasting) | 191.7 (20.34) | 188.7 (60.01) | 196.5 (48.19) | 194.2 (33.71)
  Change at Day 28: CL (fasting): number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: CL (fasting) | -9.0 (13.28) | 2.7 (15.12) | -10.8 (12.63) | 13.3 (27.09)
  Change at Day 56: CL (fasting) | 12.3 (14.19) | -10.2 (15.79) | 1.7 (12.89) | 8.0 (42.82)
  Change at Day 84: CL (fasting): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: CL (fasting) | 0.0 (8.02) | 1.5 (9.57) | -2.2 (10.80) | -2.4 (23.20)
  Change at Day 112: CL (fasting): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: CL (fasting) | -6.5 (35.23) | -5.8 (7.99) | 0.7 (19.05) | -7.2 (18.86)
  Change at Day 140: CL (fasting): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: CL (fasting) | -2.5 (17.13) | 0.3 (15.23) | 4.2 (10.67) | -5.4 (33.06)
  Change at Day 168: CL (fasting): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: CL (fasting) | -0.8 (26.54) | -2.5 (8.57) | -12.5 (21.68) | 13.0 (37.90)
  Change at Day 224/ET: CL (fasting) | -4.7 (19.79) | 0.2 (10.72) | -11.8 (24.34) | 7.2 (40.49)
  Change at Day 304/ET: CL (fasting): number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: CL (fasting) |  | 1.3 (19.28) | -3.5 (13.88) | -1.3 (29.34)
  Baseline: TG (fasting) | 141.7 (47.32) | 138.5 (58.95) | 110.5 (41.40) | 195.2 (149.85)
  Change at Day 28: TG (fasting): number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: TG (fasting) | -23.2 (35.44) | 4.0 (68.07) | -9.3 (34.91) | -8.0 (37.31)
  Change at Day 56: TG (fasting) | 4.2 (63.29) | -24.7 (57.41) | -8.2 (23.51) | -49.5 (124.64)
  Change at Day 84: TG (fasting): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: TG (fasting) | 2.2 (38.57) | -18.0 (43.32) | -19.7 (18.22) | -98.4 (140.73)
  Change at Day 112: TG (fasting): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: TG (fasting) | 6.0 (73.16) | -16.5 (32.31) | -2.8 (23.76) | -89.0 (146.53)
  Change at Day 140: TG (fasting): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: TG (fasting) | -15.0 (45.79) | -13.7 (50.39) | -7.5 (29.13) | -67.6 (84.14)
  Change at Day 168: TG (fasting): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: TG (fasting) | -11.5 (43.72) | -7.3 (26.30) | -4.2 (24.13) | -52.2 (151.28)
  Change at Day 224/ET: TG (fasting) | -24.5 (46.00) | -18.0 (54.98) | -13.8 (22.68) | -58.0 (77.36)
  Change at Day 304/ET: TG (fasting): number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: TG (fasting) |  | -18.5 (31.17) | 0.5 (26.94) | -42.0 (168.16)
  Baseline: lg G: number analyzed (Participants) | 0 | 0 | 6 | 1
  Baseline: lg G |  |  | 840.5 (171.08) | 793.0
  Change at Day 28: lg G: number analyzed (Participants) | 0 | 0 | 3 | 0
  Change at Day 28: lg G |  |  | 42.7 (26.63) |
  Change at Day 84: lg G: number analyzed (Participants) | 0 | 0 | 6 | 1
  Change at Day 84: lg G |  |  | 69.7 (65.83) | -30.0
  Change at Day 140: lg G: number analyzed (Participants) | 0 | 0 | 6 | 1
  Change at Day 140: lg G |  |  | 41.8 (72.02) | -40.0
  Baseline: lg A: number analyzed (Participants) | 0 | 0 | 6 | 1
  Baseline: lg A |  |  | 257.3 (108.27) | 299.0
  Change at Day 28: lg A: number analyzed (Participants) | 0 | 0 | 3 | 0
  Change at Day 28: lg A |  |  | 7.0 (7.55) |
  Change at Day 84: lg A: number analyzed (Participants) | 0 | 0 | 6 | 1
  Change at Day 84: lg A |  |  | -10.0 (14.56) | -25.0
  Change at Day 140: lg A: number analyzed (Participants) | 0 | 0 | 6 | 1
  Change at Day 140: lg A |  |  | -4.2 (26.36) | -25.0
  Baseline: lg M: number analyzed (Participants) | 0 | 0 | 6 | 1
  Baseline: lg M |  |  | 101.0 (60.79) | 58.0
  Change at Day 28: lg M: number analyzed (Participants) | 0 | 0 | 3 | 0
  Change at Day 28: lg M |  |  | 9.7 (8.74) |
  Change at Day 84: lg M: number analyzed (Participants) | 0 | 0 | 6 | 1
  Change at Day 84: lg M |  |  | 4.7 (7.06) | -6.0
  Change at Day 140: lg M: number analyzed (Participants) | 0 | 0 | 6 | 1
  Change at Day 140: lg M |  |  | 8.2 (19.69) | -9.0

30. Secondary Outcome: Change From Baseline in Laboratory Assessments: Protein, Albumin, Hemoglobin at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Gram per deciliter (g/dL)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Gram per deciliter (g/dL)
  Baseline: Protein | 7.07 (0.273) | 6.93 (0.273) | 6.97 (0.234) | 6.77 (0.225)
  Change at Day 28: Protein: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Protein | -0.25 (0.274) | -0.25 (0.302) | -0.23 (0.386) | -0.15 (0.266)
  Change at Day 56: Protein | -0.08 (0.392) | -0.25 (0.207) | -0.03 (0.266) | -0.10 (0.434)
  Change at Day 84: Protein: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Protein | -0.03 (0.216) | 0.02 (0.293) | 0.02 (0.407) | -0.06 (0.207)
  Change at Day 112: Protein: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Protein | -0.25 (0.339) | -0.02 (0.343) | -0.05 (0.383) | -0.06 (0.378)
  Change at Day 140: Protein: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Protein | -0.28 (0.271) | -0.17 (0.225) | -0.05 (0.259) | -0.36 (0.305)
  Change at Day 168: Protein: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Protein | -0.33 (0.273) | -0.13 (0.250) | -0.23 (0.207) | 0.00 (0.529)
  Change at Day 224/ET: Protein | -0.18 (0.354) | -0.17 (0.383) | 0.03 (0.258) | 0.35 (0.404)
  Change at Day 304/ET: Protein: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Protein |  | -0.03 (0.339) | 0.02 (0.319) | 0.10 (0.572)
  Baseline: Albumin | 4.23 (0.301) | 4.48 (0.194) | 4.43 (0.121) | 4.28 (0.172)
  Change at Day 28: Albumin: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Albumin | -0.10 (0.190) | -0.12 (0.256) | -0.13 (0.310) | -0.03 (0.175)
  Change at Day 56: Albumin | 0.08 (0.319) | -0.13 (0.151) | 0.02 (0.147) | -0.12 (0.331)
  Change at Day 84: Albumin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Albumin | 0.02 (0.098) | -0.02 (0.286) | 0.02 (0.183) | -0.06 (0.152)
  Change at Day 112: Albumin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Albumin | -0.12 (0.313) | -0.07 (0.197) | 0.02 (0.117) | -0.08 (0.277)
  Change at Day 140: Albumin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Albumin | -0.08 (0.133) | -0.15 (0.152) | 0.02 (0.232) | -0.14 (0.321)
  Change at Day 168: Albumin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Albumin | -0.17 (0.175) | -0.10 (0.155) | -0.08 (0.160) | 0.00 (0.354)
  Change at Day 224/ET: Albumin | 0.03 (0.175) | -0.05 (0.362) | -0.02 (0.075) | 0.12 (0.256)
  Change at Day 304/ET: Albumin: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Albumin |  | -0.08 (0.264) | 0.00 (0.167) | 0.13 (0.377)
  Baseline: Hemoglobin | 14.07 (1.392) | 14.28 (0.662) | 13.93 (1.007) | 13.80 (1.669)
  Change at Day 28: Hemoglobin: number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: Hemoglobin | -0.36 (0.493) | -0.38 (0.337) | -0.44 (1.029) | -0.57 (0.468)
  Change at Day 56: Hemoglobin: number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: Hemoglobin | -0.03 (0.622) | -0.68 (0.356) | 0.17 (0.308) | -0.58 (0.960)
  Change at Day 84: Hemoglobin: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: Hemoglobin | -0.28 (0.471) | 0.08 (0.576) | 0.18 (0.523) | -0.75 (0.387)
  Change at Day 112: Hemoglobin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Hemoglobin | -0.18 (0.627) | -0.12 (0.714) | -0.33 (0.905) | -0.80 (0.592)
  Change at Day 140: Hemoglobin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Hemoglobin | -0.48 (0.293) | -0.10 (0.352) | -0.25 (0.991) | -0.66 (0.581)
  Change at Day 168: Hemoglobin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Hemoglobin | -0.42 (0.462) | -0.25 (0.451) | -0.55 (0.819) | -0.58 (0.507)
  Change at Day 224/ET: Hemoglobin: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: Hemoglobin | -0.12 (0.585) | 0.00 (0.525) | 0.15 (0.709) | -0.12 (0.769)
  Change at Day 304/ET: Hemoglobin: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Hemoglobin |  | 0.28 (1.1136) | 0.05 (0.565) | -0.55 (1.473)

31. Secondary Outcome: Change From Baseline in Laboratory Assessments: Aspartate Aminotransferase, Creatine Kinase, Alanine Aminotransferase, Gamma Glutamyl Transferase (GGT), Lactate Dehydrogenase, Alkaline Phosphatase at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Description: Following parameters were analyzed for laboratory examination: Aspartate Aminotransferase (AMT), Creatine Kinase (CK), Alanine Aminotransferase (ALT), Gamma Glutamyl Transferase (GGT), Lactate Dehydrogenase (LD), Alkaline Phosphatase (AP).
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
international units per liter (IU/L)
  Baseline: AST | 22.2 (3.13) | 21.2 (1.60) | 25.5 (11.38) | 19.5 (4.55)
  Change at Day 28: AST: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: AST | -1.2 (8.16) | -1.0 (1.41) | -6.8 (12.26) | -1.3 (3.20)
  Change at Day 56: AST | 1.3 (3.93) | 0.0 (0.89) | -3.7 (10.05) | 2.5 (7.79)
  Change at Day 84: AST: number analyzed (Participants) | 6 | 6 | 6 | 4
  Change at Day 84: AST | -3.5 (2.95) | -0.2 (2.48) | -4.3 (11.02) | -0.8 (3.86)
  Change at Day 112: AST: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112: AST | 0.2 (5.81) | 2.0 (1.67) | -5.8 (11.61) | -2.2 (2.77)
  Change at Day 140: AST: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: AST | -3.3 (4.27) | -0.5 (2.35) | -5.2 (9.58) | -1.0 (4.64)
  Change at Day 168: AST: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: AST | -3.2 (2.64) | -0.3 (3.14) | -6.2 (9.26) | 0.6 (3.65)
  Change at Day 224/ET: AST | 0.3 (4.18) | -0.7 (4.27) | -3.8 (11.34) | 1.8 (2.64)
  Change at Day 304/ET: AST: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: AST |  | -0.5 (1.87) | -3.8 (9.77) | 7.5 (10.47)
  Baseline: CK | 97.2 (40.32) | 104.8 (74.79) | 80.0 (20.21) | 67.5 (26.91)
  Change at Day 28: CK: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: CK | -26.3 (26.07) | 0.7 (15.06) | -7.3 (24.10) | 9.2 (18.69)
  Change at Day 56: CK | -0.5 (79.89) | -4.2 (12.48) | 12.0 (11.45) | 8.7 (15.60)
  Change at Day 84: CK: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: CK | -15.3 (12.60) | 1.0 (18.22) | 7.5 (26.77) | 3.2 (14.20)
  Change at Day 112: CK: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112: CK | -32.5 (34.16) | 7.5 (18.73) | 2.8 (13.10) | -2.0 (19.79)
  Change at Day 140: CK: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: CK | -16.7 (28.79) | 7.7 (19.71) | 0.5 (29.92) | 53.0 (106.50)
  Change at Day 168: CK: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: CK | -29.3 (24.47) | 16.3 (45.35) | 21.7 (59.27) | 8.8 (16.16)
  Change at Day 224/ET: CK | 15.0 (43.26) | 19.0 (29.14) | 77.8 (148.91) | 7.5 (9.79)
  Change at Day 304/ET: CK: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: CK |  | 61.8 (134.00) | 19.0 (31.69) | 9.5 (8.58)
  Baseline: ALT | 17.0 (4.00) | 19.5 (1.64) | 24.3 (14.14) | 17.2 (5.27)
  Change at Day 28: ALT: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: ALT | -0.3 (5.13) | 0.3 (2.66) | -11.3 (14.24) | -0.2 (0.98)
  Change at Day 56: ALT | 1.8 (3.54) | 0.8 (1.60) | -6.2 (13.70) | 3.3 (11.24)
  Change at Day 84: ALT: number analyzed (Participants) | 6 | 6 | 6 | 4
  Change at Day 84: ALT | -1.8 (4.07) | -1.2 (2.40) | -6.8 (14.13) | -2.5 (3.32)
  Change at Day 112: ALT: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112: ALT | 8.2 (25.13) | 2.2 (2.48) | -7.2 (14.50) | -2.2 (3.96)
  Change at Day 140: ALT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: ALT | -3.0 (4.15) | -1.8 (3.49) | -6.5 (10.54) | -1.0 (4.06)
  Change at Day 168: ALT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: ALT | -2.0 (4.52) | -1.2 (3.54) | -8.7 (13.81) | 0.8 (4.55)
  Change at Day 224/ET: ALT | 1.0 (3.69) | -1.0 (3.46) | -6.7 (13.28) | 0.3 (3.44)
  Change at Day 304/ET: ALT: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: ALT |  | 0.3 (1.97) | -6.8 (12.80) | 13.8 (25.33)
  Baseline: GGT | 22.0 (6.78) | 21.5 (8.29) | 17.3 (7.37) | 20.0 (10.32)
  Change at Day 28: GGT: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: GGT | -2.7 (2.58) | -0.3 (3.93) | -1.8 (2.06) | -0.7 (1.21)
  Change at Day 56: GGT | -2.3 (3.39) | -1.3 (3.27) | 0.5 (2.59) | -0.8 (1.17)
  Change at Day 84: GGT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: GGT | -2.0 (4.05) | -0.7 (2.34) | -0.7 (4.80) | -2.0 (4.12)
  Change at Day 112: GGT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: GGT | -2.2 (6.88) | -0.8 (4.75) | -1.2 (2.48) | -1.0 (3.39)
  Change at Day 140: GGT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: GGT | -4.5 (5.01) | -2.2 (4.71) | -0.2 (2.04) | 0.0 (1.41)
  Change at Day 168: GGT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: GGT | -5.0 (4.52) | -2.3 (5.01) | -1.3 (2.73) | 0.8 (1.92)
  Change at Day 224/ET: GGT | -3.3 (3.33) | -1.5 (3.39) | 0.2 (2.56) | 1.3 (3.98)
  Change at Day 304/ET: GGT: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: GGT |  | -2.3 (4.32) | 0.5 (1.97) | 31.5 (61.07)
  Baseline: LD | 174.5 (13.40) | 174.7 (25.11) | 166.7 (19.65) | 172.0 (20.03)
  Change at Day 28: LD: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: LD | -15.7 (13.06) | -14.5 (9.89) | -8.0 (15.47) | -4.3 (20.26)
  Change at Day 56: LD: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 56: LD | -3.0 (30.42) | -10.0 (7.69) | -1.2 (13.51) | 1.2 (8.53)
  Change at Day 84: LD: number analyzed (Participants) | 6 | 6 | 6 | 4
  Change at Day 84: LD | -11.3 (9.40) | -3.5 (17.93) | -1.7 (13.69) | 3.3 (25.53)
  Change at Day 112: LD: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112: LD | -18.0 (6.90) | 0.0 (17.42) | -0.8 (12.72) | -6.0 (15.87)
  Change at Day 140: LD: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: LD | -17.3 (9.65) | -14.0 (21.95) | -1.0 (15.48) | -1.2 (16.57)
  Change at Day 168: LD: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: LD | -7.5 (18.56) | -6.5 (17.56) | -2.8 (13.51) | 0.2 (18.35)
  Change at Day 224/ET: LD | 5.7 (27.16) | -6.0 (13.11) | 4.8 (18.63) | -4.0 (18.61)
  Change at Day 304/ET: LD: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: LD |  | -5.2 (15.56) | 7.2 (19.22) | -6.5 (38.66)
  Baseline: AP | 63.5 (20.34) | 72.5 (22.65) | 59.3 (12.72) | 69.7 (9.73)
  Change at Day 28: AP: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: AP | -1.3 (3.72) | -4.0 (4.43) | -6.8 (2.50) | -1.7 (3.78)
  Change at Day 56: AP | -2.3 (6.56) | -4.7 (3.98) | -5.3 (9.87) | -0.8 (3.31)
  Change at Day 84: AP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: AP | -2.3 (8.62) | -0.8 (6.31) | -7.7 (9.67) | 0.2 (5.89)
  Change at Day 112: AP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: AP | -1.7 (7.17) | -0.5 (10.84) | -6.5 (8.24) | 5.8 (5.12)
  Change at Day 140: AP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: AP | -1.0 (12.12) | -6.5 (10.80) | -6.5 (8.98) | 1.4 (4.51)
  Change at Day 168: AP: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: AP | -1.3 (8.36) | -4.2 (10.61) | -5.8 (11.25) | 3.4 (5.55)
  Change at Day 224/ET: AP | 3.3 (9.95) | -6.0 (9.32) | -6.2 (10.94) | 8.8 (9.45)
  Change at Day 304/ET: AP: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: AP |  | -5.8 (14.80) | -3.3 (11.52) | 9.3 (18.71)

32. Secondary Outcome: Change From Baseline in Laboratory Assessments: Sodium, Potassium, Chloride, Bicarbonate, Magnesium at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Milliequivalent per liter (mEq/L)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Milliequivalent per liter (mEq/L)
  Baseline: Sodium | 140.0 (1.26) | 137.8 (5.88) | 140.0 (1.79) | 141.7 (2.07)
  Change at Day 28: Sodium: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Sodium | -2.3 (3.27) | -0.3 (4.46) | 0.3 (0.96) | -1.8 (3.43)
  Change at Day 56: Sodium | -0.3 (2.80) | 0.5 (4.97) | 0.5 (2.17) | 0.0 (2.97)
  Change at Day 84: Sodium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Sodium | -0.7 (3.01) | 1.3 (3.01) | 0.7 (3.33) | 1.2 (2.28)
  Change at Day 112: Sodium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Sodium | -0.7 (3.20) | 1.0 (3.41) | 0.7 (3.39) | 1.6 (3.13)
  Change at Day 140: Sodium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Sodium | 0.0 (1.67) | 0.0 (1.41) | 2.0 (2.45) | 1.0 (2.55)
  Change at Day 168: Sodium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Sodium | -1.3 (4.08) | 0.5 (4.14) | 3.5 (1.38) | 0.6 (3.05)
  Change at Day 224/ET: Sodium | 0.2 (2.40) | 1.5 (3.83) | 2.5 (2.07) | -0.2 (2.48)
  Change at Day 304/ET: Sodium: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Sodium |  | 1.5 (3.15) | 2.2 (2.32) | 1.0 (2.45)
  Baseline: Potassium | 4.52 (0.204) | 4.40 (0.200) | 4.22 (0.475) | 4.42 (0.354)
  Change at Day 28: Potassium: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Potassium | -0.18 (0.183) | -0.07 (0.266) | -0.08 (0.15) | -0.23 (0.427)
  Change at Day 56: Potassium | -0.18 (0.223) | -0.07 (0.266) | -0.12 (0.504) | -0.13 (0.367)
  Change at Day 84: Potassium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Potassium | -0.28 (0.248) | 0.08 (0.248) | 0.10 (0.438) | -0.16 (0.439)
  Change at Day 112: Potassium: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112: Potassium | -0.10 (0.322) | 0.10 (0.303) | 0.00 (0.490) | 0.02 (0.593)
  Change at Day 140: Potassium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Potassium | -0.20 (0.253) | 0.08 (0.160) | -0.03 (0.535) | 0.02 (0.536)
  Change at Day 168: Potassium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Potassium | 0.03 (0.121) | -0.05 (0.468) | 0.08 (0.467) | -0.04 (0.586)
  Change at Day 224/ET: Potassium | -0.20 (0.276) | 0.15 (0.394) | 0.20 (0.329) | -0.13 (0.484)
  Change at Day 304/ET: Potassium: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Potassium |  | 0.40 (0.369) | 0.38 (0.458) | -0.25 (0.173)
  Baseline: Chloride | 103.8 (2.48) | 100.8 (4.88) | 102.5 (2.66) | 104.8 (2.48)
  Change at Day 28: Chloride: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Chloride | -1.8 (2.79) | 0.7 (2.66) | 1.0 (2.71) | -1.2 (2.40)
  Change at Day 56: Chloride | -0.8 (2.40) | 1.0 (2.76) | 0.5 (2.17) | 0.2 (2.56)
  Change at Day 84: Chloride: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Chloride | -1.2 (2.48) | 0.8 (2.14) | 2.0 (3.03) | 0.6 (2.41)
  Change at Day 112: Chloride: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Chloride | -1.3 (3.72) | 0.7 (2.25) | 1.7 (2.73) | 0.8 (2.39)
  Change at Day 140: Chloride: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Chloride | -1.7 (2.88) | -0.3 (1.37) | 0.7 (1.75) | -0.2 (3.11)
  Change at Day 168: Chloride: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Chloride | -0.3 (3.83) | 1.7 (3.50) | 1.3 (1.03) | -0.6 (1.82)
  Change at Day 224/ET: Chloride | -0.3 (2.94) | 1.7 (2.34) | 0.3 (1.86) | -1.8 (3.54)
  Change at Day 304/ET: Chloride: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Chloride |  | 1.0 (1.79) | 0.5 (3.21) | -0.8 (2.99)
  Baseline: Bicarbonate | 27.0 (1.55) | 27.3 (1.03) | 26.5 (2.43) | 28.0 (1.67)
  Change at Day 28: Bicarbonate: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 28: Bicarbonate | 0.5 (2.17) | -0.7 (1.51) | -1.8 (4.15) | -1.5 (2.26)
  Change at Day 56: Bicarbonate | 1.5 (1.76) | -0.8 (1.47) | -0.5 (1.87) | -2.8 (4.12)
  Change at Day 84: Bicarbonate: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Bicarbonate | 0.7 (2.34) | -0.5 (1.87) | -1.5 (3.51) | -2.0 (2.92)
  Change at Day 112: Bicarbonate: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Bicarbonate | 1.0 (2.53) | -1.5 (0.84) | -0.7 (1.97) | -1.6 (3.51)
  Change at Day 140: Bicarbonate: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Bicarbonate | 0.3 (2.94) | -0.3 (1.21) | -0.7 (2.42) | -1.2 (2.17)
  Change at Day 168: Bicarbonate: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Bicarbonate | -0.3 (2.07) | -1.5 (2.07) | -1.2 (2.04) | -1.4 (2.07)
  Change at Day 224/ET: Bicarbonate | 0.7 (2.16) | -1.0 (2.19) | 0.2 (2.23) | -0.8 (3.43)
  Change at Day 304/ET: Bicarbonate: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Bicarbonate |  | 0.2 (3.06) | -1.5 (1.64) | -1.0 (2.94)
  Baseline: Magnesium | 1.72 (0.075) | 1.88 (0.160) | 1.67 (0.294) | 1.83 (0.052)
  Change at Day 28: Magnesium: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: Magnesium | 0.03 (0.052) | -0.03 (0.103) | -0.02 (0.126) | -0.10 (0.000)
  Change at Day 56: Magnesium | -0.03 (0.082) | -0.05 (0.138) | -0.02 (0.133) | 0.00 (0.063)
  Change at Day 84: Magnesium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Magnesium | 0.00 (0.089) | 0.03 (0.151) | 0.03 (0.082) | 0.00 (0.122)
  Change at Day 112: Magnesium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Magnesium | 0.02 (0.075) | 0.02 (0.160) | 0.05 (0.084) | -0.02 (0.084)
  Change at Day 140: Magnesium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Magnesium | 0.02 (0.075) | -0.05 (0.176) | -0.03 (0.082) | -0.06 (0.055)
  Change at Day 168: Magnesium: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Magnesium | -0.02 (0.098) | 0.00 (0.200) | -0.05 (0.055) | -0.02 (0.130)
  Change at Day 224/ET: Magnesium | -0.02 (0.098) | 0.00 (0.126) | -0.03 (0.103) | -0.07 (0.121)
  Change at Day 304/ET: Magnesium: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Magnesium |  | -0.02 (0.147) | 0.00 (0.089) | -0.10 (0.183)

33. Secondary Outcome: Change From Baseline in Laboratory Assessments: Hematocrit at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Description: Following hematology parameters were analyzed for laboratory examination: Hemoglobin, Hematocrit, Red blood cell (RBC) count, Platelet count, WBC count, Total neutrophils (Abs),Eosinophils (Abs),Monocytes (Abs),Basophils (Abs), Lymphocytes (Abs).
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of RBCs to total blood volume
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Percentage of RBCs to total blood volume
  Baseline: Hematocrit | 41.70 (3.906) | 41.28 (2.436) | 40.78 (2.927) | 40.87 (5.369)
  Change at Day 28: Hematocrit: number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: Hematocrit | -1.18 (1.161) | -0.67 (0.864) | -1.28 (3.342) | -1.73 (1.866)
  Change at Day 56: Hematocrit: number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: Hematocrit | -0.25 (1.545) | -1.68 (0.823) | 0.90 (0.876) | -1.35 (2.914)
  Change at Day 84: Hematocrit: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: Hematocrit | -0.53 (1.458) | 0.56 (1.593) | 1.25 (1.714) | -1.85 (1.771)
  Change at Day 112: Hematocrit: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 112: Hematocrit | 0.07 (2.272) | 0.08 (2.464) | -0.34 (3.140) | -2.18 (1.847)
  Change at Day 140: Hematocrit: number analyzed (Participants) | 6 | 6 | 6 | 4
  Change at Day 140: Hematocrit | -0.60 (1.797) | 0.53 (1.280) | -0.78 (2.920) | -1.30 (1.687)
  Change at Day 168: Hematocrit: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Hematocrit | -1.47 (1.480) | 0.05 (1.294) | -1.20 (3.251) | -1.26 (0.730)
  Change at Day 224/ET: Hematocrit: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: Hematocrit | -0.30 (1.611) | 1.50 (1.745) | 1.15 (2.393) | 0.22 (2.845)
  Change at Day 304/ET: Hematocrit: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Hematocrit |  | 2.07 (3.841) | 0.23 (2.007) | -1.10 (5.412)

34. Secondary Outcome: Change From Baseline in Laboratory Assessments: Red Blood Cells (RBCs) at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliter
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
10^6 cells/microliter
  Baseline: RBC | 4.45 (0.394) | 4.48 (0.407) | 4.42 (0.417) | 4.43 (0.677)
  Change at Day 28: RBC: number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: RBC | -0.10 (0.141) | -0.07 (0.103) | -0.14 (0.358) | -0.15 (0.176)
  Change at Day 56: RBC: number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: RBC | 0.02 (0.160) | -0.18 (0.110) | 0.02 (0.098) | -0.10 (0.335)
  Change at Day 84: RBC: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: RBC | -0.03 (0.151) | 0.00 (0.255) | 0.07 (0.121) | -0.23 (0.126)
  Change at Day 112: RBC: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: RBC | 0.03 (0.207) | -0.05 (0.302) | -0.13 (0.242) | -0.22 (0.277)
  Change at Day 140: RBC: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: RBC | -0.07 (0.207) | -0.03 (0.207) | -0.13 (0.333) | -0.08 (0.277)
  Change at Day 168: RBC: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: RBC | -0.12 (0.172) | -0.03 (0.163) | -0.22 (0.319) | -0.10 (0.187)
  Change at Day 224/ET: RBC: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: RBC | -0.02 (0.160) | 0.10 (0.110) | 0.03 (0.320) | 0.00 (0.292)
  Change at Day 304/ET: RBC: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: RBC |  | 0.15 (0.442) | -0.02 (0.214) | -0.23 (0.443)

35. Secondary Outcome: Change From Baseline in Laboratory Assessments: Platelets, White Blood Cells (WBCs), Neutrophils (Absolute), Eosinophils (Absolute), Basophils (Absolute), Lymphocytes (Absolute), Monocytes (Absolute) at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
10^3 cells/microliter
  Baseline: Platelets | 187.5 (50.91) | 209.3 (39.52) | 198.7 (57.30) | 204.2 (51.86)
  Change at Day 28: Platelets: number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: Platelets | 1.2 (13.55) | -10.7 (21.99) | -7.0 (22.30) | 0.7 (17.19)
  Change at Day 56: Platelets: number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: Platelets | -1.0 (15.38) | -14.4 (24.27) | 9.3 (14.49) | -3.2 (18.85)
  Change at Day 84: Platelets: number analyzed (Participants) | 5 | 5 | 6 | 4
  Change at Day 84: Platelets | -0.6 (14.17) | 4.0 (22.90) | -1.0 (11.54) | 9.8 (31.96)
  Change at Day 112: Platelets: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Platelets | 13.5 (21.19) | -3.5 (31.05) | 27.3 (55.97) | 10.4 (29.95)
  Change at Day 140: Platelets: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Platelets | 5.2 (20.97) | -12.2 (16.80) | -2.7 (41.86) | -2.0 (17.72)
  Change at Day 168: Platelets: number analyzed (Participants) | 6 | 5 | 5 | 5
  Change at Day 168: Platelets | 4.5 (26.16) | -1.2 (28.49) | 5.2 (13.52) | -2.0 (35.94)
  Change at Day 224/ET: Platelets: number analyzed (Participants) | 5 | 6 | 6 | 5
  Change at Day 224/ET: Platelets | 5.4 (9.56) | -5.5 (27.29) | 19.3 (30.32) | 0.2 (24.77)
  Change at Day 304/ET: Platelets: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Platelets |  | -11.8 (30.33) | 15.5 (16.36) | 6.0 (37.05)
  Baseline: WBC | 5.75 (1.744) | 6.08 (1.023) | 6.17 (1.334) | 7.40 (2.497)
  Change at Day 28: WBC: number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: WBC | -0.02 (1.163) | -0.40 (0.839) | -0.54 (0.783) | -1.02 (1.880)
  Change at Day 56: WBC: number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: WBC | 0.15 (1.104) | -0.42 (0.676) | -0.07 (0.579) | -1.75 (1.260)
  Change at Day 84: WBC: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: WBC | 0.30 (1.410) | -0.28 (1.326) | -0.33 (0.463) | -1.08 (1.721)
  Change at Day 112: WBC: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: WBC | 0.05 (1.048) | 0.32 (1.341) | -0.35 (1.417) | -0.76 (1.408)
  Change at Day 140: WBC: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: WBC | -0.33 (1.414) | 0.03 (1.166) | -0.87 (1.571) | -1.06 (1.324)
  Change at Day 168: WBC: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: WBC | -0.08 (1.280) | -0.13 (1.657) | -0.82 (0.454) | -0.16 (1.766)
  Change at Day 224/ET: WBC: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: WBC | 0.35 (1.693) | -0.42 (0.882) | -0.10 (0.395) | -0.82 (1.329)
  Change at Day 304/ET: WBC: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: WBC |  | -0.18 (1.743) | 0.60 (2.199) | -0.98 (1.513)
  Baseline: Neutrophils (abs) | 3.508 (1.4359) | 3.813 (1.1002) | 3.637 (0.8430) | 5.077 (2.3807)
  Change at Day 28: Neutrophils (abs): number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: Neutrophils (abs) | 0.154 (0.8442) | -0.320 (0.7102) | -0.264 (0.4348) | -0.730 (1.9961)
  Change at Day 56: Neutrophils (abs): number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: Neutrophils (abs) | 0.237 (1.1972) | -0.226 (0.7418) | -0.007 (0.4337) | -1.342 (1.2706)
  Change at Day 84: Neutrophils (abs): number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: Neutrophils (abs) | 0.405 (1.3205) | -0.062 (0.9878) | -0.100 (0.3685) | -0.925 (1.7647)
  Change at Day 112: Neutrophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Neutrophils (abs) | 0.043 (0.8887) | 0.455 (1.2804) | 0.218 (1.3491) | -0.502 (1.5264)
  Change at Day 140: Neutrophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Neutrophils (abs) | -0.348 (1.1549) | 0.260 (1.1844) | -0.313 (1.3322) | -0.968 (1.6410)
  Change at Day 168: Neutrophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Neutrophils (abs) | 0.137 (0.9677) | 0.092 (1.5919) | -0.398 (0.3572) | -0.020 (1.9093)
  Change at Day 224/ET: Neutrophils(abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: Neutrophils(abs) | 0.413 (1.3356) | -0.188 (0.7241) | 0.088 (0.4068) | -0.972 (1.1744)
  Change at Day 304/ET: Neutrophils(abs): number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Neutrophils(abs) |  | -0.035 (1.3786) | 0.838 (1.8792) | -0.815 (1.3199)
  Baseline: Eosinophils (abs) | 0.212 (0.1298) | 0.242 (0.0823) | 0.208 (0.1338) | 0.162 (0.1005)
  Change at Day 28: Eosinophils (abs): number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: Eosinophils (abs) | 0.012 (0.0638) | 0.020 (0.0994) | 0.012 (0.0676) | 0.027 (0.0871)
  Change at Day 56: Eosinophils (abs): number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: Eosinophils (abs) | -0.002 (0.0898) | 0.012 (0.1215) | 0.017 (0.0909) | -0.007 (0.0628)
  Change at Day 84: Eosinophils (abs): number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: Eosinophils (abs) | -0.007 (0.0547) | 0.074 (0.0832) | -0.008 (0.0643) | 0.043 (0.0842)
  Change at Day 112: Eosinophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Eosinophils (abs) | -0.008 (0.0685) | 0.053 (0.1285) | -0.045 (0.0547) | 0.058 (0.1003)
  Change at Day 140: Eosinophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Eosinophils (abs) | 0.028 (0.0567) | -0.005 (0.0892) | -0.078 (0.0652) | 0.032 (0.0750)
  Change at Day 168: Eosinophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Eosinophils (abs) | -0.042 (0.0786) | 0.012 (0.0467) | -0.082 (0.0891) | 0.030 (0.0903)
  Change at Day 224/ET: Eosinophils(abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: Eosinophils(abs) | -0.015 (0.0740) | 0.002 (0.0830) | -0.057 (0.0831) | 0.076 (0.1328)
  Change at Day 304/ET: Eosinophils(abs): number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Eosinophils(abs) |  | -0.010 (0.1122) | -0.010 (0.0447) | 0.075 (0.1318)
  Baseline: Basophils (abs) | 0.032 (0.0133) | 0.048 (0.0371) | 0.032 (0.0214) | 0.030 (0.0200)
  Change at Day 28: Basophils (abs): number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: Basophils (abs) | 0.014 (0.0358) | -0.012 (0.0549) | 0.002 (0.0349) | -0.003 (0.0258)
  Change at Day 56: Basophils (abs): number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: Basophils (abs) | 0.003 (0.0137) | -0.016 (0.0611) | 0.008 (0.0214) | -0.005 (0.0176)
  Change at Day 84: Basophils (abs): number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: Basophils (abs) | 0.007 (0.0175) | -0.014 (0.0404) | -0.008 (0.0204) | 0.000 (0.0216)
  Change at Day 112: Basophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Basophils (abs) | 0.003 (0.0103) | -0.022 (0.0422) | 0.008 (0.0194) | 0.002 (0.0217)
  Change at Day 140: Basophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Basophils (abs) | 0.003 (0.0137) | -0.027 (0.0344) | -0.003 (0.0225) | 0.000 (0.0265)
  Change at Day 168: Basophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Basophils (abs) | 0.005 (0.0266) | -0.025 (0.0378) | -0.007 (0.0225) | 0.022 (0.0363)
  Change at Day 224/ET: Basophils (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: Basophils (abs) | -0.008 (0.0147) | -0.027 (0.0294) | 0.007 (0.0378) | 0.012 (0.0179)
  Change at Day 304/ET: Basophils (abs): number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Basophils (abs) |  | -0.028 (0.0223) | -0.012 (0.0256) | 0.010 (0.0082)
  Baseline: Lymphocytes (abs) | 1.470 (0.3329) | 1.528 (0.3669) | 1.748 (0.4477) | 1.598 (0.3810)
  Change at Day 28: Lymphocytes (abs): number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: Lymphocytes (abs) | -0.160 (0.2853) | -0.088 (0.2491) | -0.198 (0.1997) | -0.197 (0.3760)
  Change at Day 56: Lymphocytes (abs): number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: Lymphocytes (abs) | -0.042 (0.1594) | -0.190 (0.2155) | 0.023 (0.2467) | -0.273 (0.3223)
  Change at Day 84: Lymphocytes (abs): number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: Lymphocytes (abs) | -0.063 (0.1973) | -0.256 (0.4282) | -0.090 (0.1452) | -0.108 (0.0171)
  Change at Day 112: Lymphocytes (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Lymphocytes (abs) | 0.023 (0.2299) | -0.145 (0.3142) | -0.303 (0.2717) | -0.238 (0.3872)
  Change at Day 140: Lymphocytes (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Lymphocytes (abs) | 0.012 (0.2175) | -0.188 (0.2584) | -0.293 (0.0907) | -0.084 (0.4824)
  Change at Day 168: Lymphocytes (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Lymphocytes (abs) | -0.173 (0.2486) | -0.192 (0.1985) | -0.192 (0.2218) | -0.152 (0.5413)
  Change at Day 224/ET: Lymphocytes(abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: Lymphocytes(abs) | -0.025 (0.3961) | -0.200 (0.1579) | -0.048 (0.2303) | 0.118 (0.3841)
  Change at Day 304/ET: Lymphocytes(abs): number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Lymphocytes(abs) |  | -0.128 (0.2971) | -0.180 (0.3600) | -0.180 (0.1911)
  Baseline: Monocytes (abs) | 0.522 (0.1622) | 0.455 (0.1440) | 0.525 (0.1169) | 0.542 (0.1569)
  Change at Day 28: Monocytes (abs): number analyzed (Participants) | 5 | 6 | 5 | 6
  Change at Day 28: Monocytes (abs) | -0.034 (0.1826) | -0.033 (0.0898) | -0.084 (0.0899) | -0.127 (0.1488)
  Change at Day 56: Monocytes (abs): number analyzed (Participants) | 6 | 5 | 6 | 6
  Change at Day 56: Monocytes (abs) | -0.043 (0.1229) | -0.020 (0.0265) | -0.095 (0.0517) | -0.133 (0.1402)
  Change at Day 84: Monocytes (abs): number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: Monocytes (abs) | -0.040 (0.1185) | -0.022 (0.0991) | -0.102 (0.0700) | -0.100 (0.0702)
  Change at Day 112: Monocytes (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Monocytes (abs) | 0.000 (0.0701) | -0.017 (0.1061) | -0.203 (0.1183) | -0.090 (0.0620)
  Change at Day 140: Monocytes (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Monocytes (abs) | -0.020 (0.1753) | -0.013 (0.1058) | -0.177 (0.2366) | -0.068 (0.1283)
  Change at Day 168: Monocytes (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: Monocytes (abs) | -0.005 (0.1566) | -0.017 (0.1216) | -0.128 (0.0781) | -0.080 (0.0718)
  Change at Day 224/ET: Monocytes (abs): number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 224/ET: Monocytes (abs) | -0.023 (0.1649) | -0.025 (0.1154) | -0.077 (0.0789) | -0.080 (0.1259)
  Change at Day 304/ET: Monocytes (abs): number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Monocytes (abs) |  | 0.012 (0.1620) | -0.017 (0.1188) | -0.065 (0.0915)

36. Secondary Outcome: Change From Baseline in Laboratory Assessments: Prothrombin Time (PT), Partial Thromboplastin Time at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Description: Following hematology parameters were analyzed for laboratory examination: Prothrombin Time (PT), Partial Thromboplastin Time.
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Second
  Baseline: PT | 11.82 (0.556) | 11.53 (0.505) | 11.10 (1.056) | 11.90 (1.220)
  Change at Day 28: PT: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 28: PT | -0.55 (0.362) | -0.02 (0.248) | 0.18 (0.896) | -0.58 (1.143)
  Change at Day 56: PT: number analyzed (Participants) | 5 | 6 | 5 | 4
  Change at Day 56: PT | 0.10 (0.758) | -0.28 (0.920) | 0.12 (0.766) | -0.27 (2.025)
  Change at Day 84: PT: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: PT | -0.25 (0.327) | -0.12 (0.676) | 0.37 (1.221) | -0.95 (1.353)
  Change at Day 112: PT: number analyzed (Participants) | 5 | 6 | 5 | 4
  Change at Day 112: PT | 0.20 (1.259) | -0.43 (0.308) | 0.60 (1.356) | -1.00 (1.383)
  Change at Day 140: PT: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 140: PT | 0.47 (0.700) | 0.17 (0.802) | 0.24 (0.820) | -0.26 (2.019)
  Change at Day 168: PT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: PT | -0.32 (1.326) | -0.37 (0.871) | 0.15 (0.609) | -0.80 (1.037)
  Change at Day 224/ET: PT | -0.67 (0.931) | -0.42 (0.407) | -0.28 (0.783) | -0.77 (1.510)
  Change at Day 304/ET: PT: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: PT |  | -0.05 (0.750) | -0.73 (0.528) | -0.42 (2.050)
  Baseline: PTT | 31.12 (3.842) | 32.57 (4.457) | 31.63 (6.808) | 31.23 (5.460)
  Change at Day 28: PTT: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 28: PTT | -1.77 (4.431) | -0.33 (1.490) | -3.86 (5.106) | 0.17 (2.521)
  Change at Day 56: PTT: number analyzed (Participants) | 5 | 6 | 5 | 4
  Change at Day 56: PTT | -4.64 (7.314) | 0.45 (2.338) | -1.00 (7.216) | -0.52 (3.801)
  Change at Day 84: PTT: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: PTT | -3.08 (4.275) | 0.44 (2.235) | 1.73 (12.794) | 0.00 (2.302)
  Change at Day 112: PTT: number analyzed (Participants) | 5 | 6 | 5 | 4
  Change at Day 112: PTT | -0.18 (6.184) | -2.42 (2.870) | 1.06 (5.949) | -0.02 (1.424)
  Change at Day 140: PTT: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 140: PTT | 0.18 (5.651) | -2.02 (1.105) | 0.22 (6.524) | -2.02 (2.751)
  Change at Day 168: PTT: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: PTT | -1.83 (4.898) | -0.48 (3.284) | 2.78 (8.713) | -0.52 (2.840)
  Change at Day 224/ET: PTT | -2.47 (3.686) | 0.90 (4.901) | 1.68 (6.563) | -0.28 (2.869)
  Change at Day 304/ET: PTT: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: PTT |  | 1.92 (3.381) | 4.83 (5.654) | 3.95 (8.973)

37. Secondary Outcome: Change From Baseline in Laboratory Assessments: Urine Specific Gravity at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Description: Urine specific gravity is a measure of the ratio of the density of urine to the density of water.
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
ratio
  Baseline: USG | 1.0197 (0.00565) | 1.0150 (0.00529) | 1.0138 (0.00343) | 1.0242 (0.00615)
  Change at Day 28: USG: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 28: USG | -0.0018 (0.00950) | 0.0012 (0.00462) | 0.0020 (0.00636) | -0.0043 (0.00383)
  Change at Day 56: USG | -0.0018 (0.00741) | -0.0003 (0.00787) | 0.0022 (0.00293) | -0.0025 (0.00259)
  Change at Day 84: USG: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: USG | -0.0010 (0.00654) | -0.0008 (0.00376) | -0.0002 (0.00293) | -0.0020 (0.00474)
  Change at Day 112: USG: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: USG | -0.0010 (0.00940) | -0.0005 (0.00625) | 0.0047 (0.00680) | 0.0002 (0.00277)
  Change at Day 140: USG: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: USG | -0.0002 (0.00462) | -0.0020 (0.00447) | 0.0015 (0.00650) | -0.0022 (0.00492)
  Change at Day 168: USG: number analyzed (Participants) | 6 | 5 | 6 | 5
  Change at Day 168: USG | 0.0008 (0.00884) | -0.0012 (0.00559) | 0.0045 (0.00568) | -0.0024 (0.00493)
  Change at Day 224/ET: USG | -0.0013 (0.00266) | -0.0003 (0.00497) | 0.0038 (0.00366) | -0.0022 (0.00527)
  Change at Day 304/ET: USG: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: USG |  | -0.0028 (0.00768) | 0.0058 (0.00591) | -0.0010 (0.00566)

38. Secondary Outcome: Change From Baseline in Laboratory Assessments: Urine pH at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Description: Urine pH is a method for evaluating urine acidity measured on a 10-point scale ranging from 0 (most acidic) to 9 (most alkaline). A lower pH means more acidity.
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
units on a scale
  Baseline: Urine pH | 6.33 (0.408) | 5.92 (0.376) | 6.00 (0.000) | 6.00 (0.316)
  Change at Day 28: Urine pH: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 28: Urine pH | -0.17 (0.258) | 0.42 (0.376) | 0.30 (0.447) | -0.08 (0.492)
  Change at Day 56: Urine pH | 0.00 (0.447) | 0.17 (0.408) | 0.08 (0.204) | 0.08 (0.585)
  Change at Day 84: Urine pH: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 84: Urine pH | -0.08 (0.376) | 0.00 (0.447) | 0.25 (0.524) | 0.20 (0.274)
  Change at Day 112: Urine pH: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 112: Urine pH | 0.08 (0.585) | 0.00 (0.316) | 0.17 (0.408) | -0.20 (0.570)
  Change at Day 140: Urine pH: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 140: Urine pH | -0.25 (0.274) | 0.50 (0.548) | 0.25 (0.524) | 0.00 (0.500)
  Change at Day 168: Urine pH: number analyzed (Participants) | 6 | 5 | 6 | 5
  Change at Day 168: Urine pH | -0.08 (0.492) | 0.30 (0.671) | 0.17 (0.516) | 0.00 (0.354)
  Change at Day 224/ET: Urine pH | -0.17 (0.408) | 0.25 (0.689) | 0.75 (0.935) | -0.17 (0.258)
  Change at Day 304/ET: Urine pH: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: Urine pH |  | 0.33 (0.408) | 0.25 (0.418) | -0.13 (0.479)

39. Secondary Outcome: Change From Baseline in Laboratory Assessments: Beta Interleukin-1, Interleukin-6, Alpha Tumor Necrosis Factor, Interferon (Gamma) at Day 28, 56, 84, 112, 140
Time Frame: Baseline, Day 28, 56, 84, 112, 140
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Picogram per milliliter (pg/ml)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Picogram per milliliter (pg/ml)
  Baseline: beta IL-1: number analyzed (Participants) | 6 | 0 | 0 | 2
  Baseline: beta IL-1 | 0.00 (0.000) |  |  | 0.00 (0.000)
  Change at Day 28: beta IL-1: number analyzed (Participants) | 6 | 0 | 0 | 2
  Change at Day 28: beta IL-1 | 0.32 (0.776) |  |  | 0.00 (0.000)
  Change at Day 56: beta IL-1: number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 56: beta IL-1 | 0.00 (0.000) |  |  | 0.00
  Change at Day 84: beta IL-1: number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 84: beta IL-1 | 0.40 (0.980) |  |  | 0.00
  Change at Day 112: beta IL-1: number analyzed (Participants) | 5 | 0 | 0 | 1
  Change at Day 112: beta IL-1 | 0.00 (0.000) |  |  | 0.00
  Change at Day 140: beta IL-1: number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 140: beta IL-1 | 0.23 (0.572) |  |  | 0.00
  Baseline: IL-6: number analyzed (Participants) | 6 | 6 | 6 | 5
  Baseline: IL-6 | 0.00 (0.000) | 1.22 (1.354) | 0.62 (1.511) | 0.52 (1.163)
  Change at Day 28: IL-6: number analyzed (Participants) | 6 | 6 | 4 | 5
  Change at Day 28: IL-6 | 0.90 (1.445) | -1.22 (1.354) | 1.23 (4.190) | 0.34 (0.760)
  Change at Day 56: IL-6: number analyzed (Participants) | 6 | 6 | 4 | 4
  Change at Day 56: IL-6 | 0.67 (1.633) | -1.22 (1.354) | 0.10 (3.186) | 0.20 (0.400)
  Change at Day 84: IL-6: number analyzed (Participants) | 6 | 4 | 6 | 4
  Change at Day 84: IL-6 | 0.00 (0.000) | 1.50 (2.386) | -0.05 (2.247) | 0.50 (1.000)
  Change at Day 112: IL-6: number analyzed (Participants) | 5 | 6 | 6 | 4
  Change at Day 112: IL-6 | 1.84 (2.855) | -0.05 (2.002) | -0.62 (1.511) | 0.55 (1.168)
  Change at Day 140: IL-6: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 140: IL-6 | 0.00 (0.000) | 0.90 (3.366) | 3.38 (5.754) | 1.63 (1.950)
  Baseline: alpha TNF: number analyzed (Participants) | 6 | 0 | 0 | 2
  Baseline: alpha TNF | 2.943 (1.7942) |  |  | 3.185 (1.2657)
  Change at Day 28: alpha TNF: number analyzed (Participants) | 6 | 0 | 0 | 2
  Change at Day 28: alpha TNF | 1.175 (2.0170) |  |  | -1.425 (1.2233)
  Change at Day 56: alpha TNF: number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 56: alpha TNF | 0.590 (2.2536) |  |  | 0.790
  Change at Day 84: alpha TNF: number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 84: alpha TNF | 1.423 (1.2367) |  |  | 0.520
  Change at Day 112: alpha TNF: number analyzed (Participants) | 5 | 0 | 0 | 1
  Change at Day 112: alpha TNF | 1.762 (1.5999) |  |  | 1.140
  Change at Day 140: alpha TNF: number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 140: alpha TNF | 1.512 (1.4736) |  |  | 1.220
  Baseline: INF (Gamma): number analyzed (Participants) | 6 | 0 | 0 | 2
  Baseline: INF (Gamma) | 0.0 (0.00) |  |  | 0.0 (0.00)
  Change at Day 28: INF (Gamma): number analyzed (Participants) | 6 | 0 | 0 | 2
  Change at Day 28: INF (Gamma) | 0.0 (0.00) |  |  | 0.0 (0.00)
  Change at Day 56: INF (Gamma): number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 56: INF (Gamma) | 0.0 (0.00) |  |  | 0.0
  Change at Day 84: INF (Gamma): number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 84: INF (Gamma) | 0.0 (0.00) |  |  | 0.0
  Change at Day 112: INF (Gamma): number analyzed (Participants) | 5 | 0 | 0 | 1
  Change at Day 112: INF (Gamma) | 0.0 (0.00) |  |  | 0.0
  Change at Day 140: INF (Gamma): number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 140: INF (Gamma) | 0.0 (0.00) |  |  | 0.0

40. Secondary Outcome: Change From Baseline in Laboratory Assessments: Component of Complement (C3A, C5B-9) at Day 28, 56, 84, 112, 140
Time Frame: Baseline, Day 28, 56, 84, 112, 140
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Nanogram per milliliter (ng/mL)
  Baseline: C3A | 970.3 (214.77) | 928.0 (228.37) | 1465.8 (352.95) | 1813.0 (1060.66)
  Change at Day 28: C3A: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: C3A | 560.2 (1109.51) | 447.5 (457.21) | 161.3 (523.83) | -305.3 (899.05)
  Change at Day 56: C3A ): number analyzed (Participants) | 6 | 6 | 4 | 5
  Change at Day 56: C3A ) | 404.7 (280.70) | 221.0 (202.67) | -74.5 (723.41) | -220.6 (231.43)
  Change at Day 84: C3A: number analyzed (Participants) | 6 | 5 | 6 | 5
  Change at Day 84: C3A | 380.3 (341.07) | 290.2 (414.07) | -610.3 (425.31) | 117.0 (826.44)
  Change at Day 112: C3A: number analyzed (Participants) | 5 | 6 | 6 | 5
  Change at Day 112: C3A | 445.2 (465.87) | 246.0 (337.86) | -129.5 (454.93) | 746.2 (1686.03)
  Change at Day 140: C3A: number analyzed (Participants) | 6 | 5 | 6 | 5
  Change at Day 140: C3A | 297.8 (508.62) | 928.6 (398.79) | -68.3 (543.15) | -32.2 (846.33)
  Baseline: C5B-9 | 289.5 (56.64) | 199.8 (16.87) | 244.3 (132.87) | 299.7 (154.14)
  Change at Day 28: C5B-9: number analyzed (Participants) | 6 | 6 | 4 | 6
  Change at Day 28: C5B-9 | -33.5 (83.69) | -26.2 (44.51) | -63.0 (131.56) | -85.5 (87.54)
  Change at Day 56: C5B-9: number analyzed (Participants) | 6 | 6 | 4 | 5
  Change at Day 56: C5B-9 | -78.0 (47.76) | 11.3 (59.09) | 0.0 (50.73) | -8.0 (109.90)
  Change at Day 84: C5B-9: number analyzed (Participants) | 6 | 5 | 6 | 5
  Change at Day 84: C5B-9 | -9.8 (152.15) | 16.6 (105.20) | 34.5 (102.80) | 4.8 (86.14)
  Change at Day 112: C5B-9: number analyzed (Participants) | 5 | 6 | 6 | 5
  Change at Day 112: C5B-9 | -35.8 (63.01) | -15.3 (36.68) | 51.8 (106.84) | 42.6 (99.64)
  Change at Day 140: C5B-9: number analyzed (Participants) | 6 | 5 | 6 | 5
  Change at Day 140: C5B-9 | -36.8 (69.42) | -10.2 (123.29) | -13.3 (98.95) | -30.2 (74.25)

41. Secondary Outcome: Change From Baseline in Laboratory Assessments: Cluster of Differentiation 4 (C4D) at Day 28, 56, 84, 112, 140
Time Frame: Baseline, Day 28, 56, 84, 112, 140
Population: All randomized participants who met the inclusion criteria and received any amount of study drug were included. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluated for given time point.
Measure: Mean (Standard Deviation); unit: Microgram per milliliter (mcg/mL)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 0 | 0 | 6
Microgram per milliliter (mcg/mL)
  Baseline: C4D: number analyzed (Participants) | 6 | 0 | 0 | 2
  Baseline: C4D | 2.692 (1.5264) |  |  | 3.720 (2.2910)
  Change at Day 28: C4D: number analyzed (Participants) | 6 | 0 | 0 | 2
  Change at Day 28: C4D | 1.078 (4.3643) |  |  | -1.720 (1.0748)
  Change at Day 56: C4D: number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 56: C4D | -1.503 (1.4911) |  |  | -1.320
  Change at Day 84: C4D: number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 84: C4D | -0.907 (1.6772) |  |  | 1.180
  Change at Day 112: C4D: number analyzed (Participants) | 5 | 0 | 0 | 1
  Change at Day 112: C4D | -0.466 (1.6322) |  |  | 1.060
  Change at Day 140: C4D: number analyzed (Participants) | 6 | 0 | 0 | 1
  Change at Day 140: C4D | -0.338 (1.6790) |  |  | 0.140

42. Secondary Outcome: Change From Baseline in Prothrombin Time (PT) International Normalized Ratio (INR) at Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Time Frame: Baseline, Day 28, 56, 84, 112, 140, 168, 224, 304/ET
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Ratio
  Baseline: PT-INR | 0.995 (0.0455) | 0.972 (0.0436) | 0.933 (0.0871) | 1.017 (0.1167)
  Change at Day 28: PT-INR: number analyzed (Participants) | 6 | 6 | 5 | 6
  Change at Day 28: PT-INR | -0.047 (0.0288) | -0.003 (0.0234) | 0.064 (0.1199) | -0.050 (0.0925)
  Change at Day 56: PT-INR: number analyzed (Participants) | 5 | 6 | 5 | 4
  Change at Day 56: PT-INR | 0.006 (0.0586) | -0.027 (0.0755) | 0.096 (0.0623) | 0.000 (0.1802)
  Change at Day 84: PT-INR: number analyzed (Participants) | 6 | 5 | 6 | 4
  Change at Day 84: PT-INR | -0.022 (0.0256) | 0.004 (0.0522) | 0.117 (0.1076) | -0.060 (0.1374)
  Change at Day 112: PT-INR: number analyzed (Participants) | 5 | 6 | 5 | 4
  Change at Day 112: PT-INR | 0.014 (0.1001) | -0.008 (0.0488) | 0.140 (0.1231) | -0.062 (0.1284)
  Change at Day 140: PT-INR: number analyzed (Participants) | 6 | 6 | 5 | 5
  Change at Day 140: PT-INR | 0.037 (0.0535) | 0.042 (0.0697) | 0.106 (0.0669) | -0.006 (0.1757)
  Change at Day 168: PT-INR: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: PT-INR | -0.027 (0.1078) | -0.005 (0.0912) | 0.098 (0.0519) | -0.050 (0.1077)
  Change at Day 224/ET: PT-INR | -0.058 (0.0776) | 0.047 (0.0344) | 0.060 (0.0651) | -0.018 (0.1148)
  Change at Day 304/ET: PT-INR: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: PT-INR |  | 0.085 (0.0599) | 0.055 (0.0481) | 0.050 (0.1927)

43. Secondary Outcome: Change From Electrocardiogram (ECG): QTcF Interval (Fridericia's Correction) at Day 1, 28, 56, 84, 112, 140, 168, 224, 304/ET
Description: QT interval corrected using the Fridericia formula (QTcF) >=500 msec; Maximum Change from Baseline in QTcF at Borderline >=30 msec to <60 msec and Prolonged >=60 msec.
Time Frame: as for outcome 27
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Millisecond (msec)
  Baseline: QTcF | 414.22 (13.474) | 427.89 (21.462) | 420.56 (20.579) | 412.06 (20.201)
  Change at 1 H post-dose Day 1: QTcF | 0.56 (8.035) | -1.50 (4.732) | 3.06 (8.762) | 3.86 (13.329)
  Change at 4 H post-dose Day 1: QTcF | 1.50 (14.898) | -8.78 (13.480) | 1.50 (13.328) | 9.50 (28.659)
  Change at pre-dose Day 28: QTcF | -4.72 (15.874) | -12.06 (14.565) | 1.78 (15.022) | -2.06 (8.410)
  Change at pre-dose Day 56: QTcF | -2.22 (13.404) | -6.06 (9.799) | 7.11 (19.452) | 6.44 (15.930)
  Change at pre-dose Day 84: QTcF: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 84: QTcF | -1.39 (10.438) | -9.72 (14.220) | 6.11 (20.435) | 19.00 (24.226)
  Change at pre-dose Day 112: QTcF: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 112: QTcF | -5.22 (8.005) | -5.89 (10.681) | 0.78 (8.275) | 25.80 (39.012)
  Change at pre-dose Day 140: QTcF: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at pre-dose Day 140: QTcF | -2.67 (7.598) | -0.11 (8.614) | 8.61 (7.672) | 8.87 (23.092)
  Change at 1 H post-dose Day 140: QTcF: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 1 H post-dose Day 140: QTcF | -2.28 (9.488) | -15.83 (36.907) | 10.61 (11.174) | 14.13 (15.604)
  Change at 4 H post dose Day 140: QTcF: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at 4 H post dose Day 140: QTcF | -3.17 (7.001) | -3.28 (8.510) | 12.72 (8.172) | 11.60 (19.991)
  Change at Day 168: QTcF: number analyzed (Participants) | 6 | 6 | 6 | 5
  Change at Day 168: QTcF | -8.56 (16.363) | -1.22 (12.523) | 7.94 (18.671) | 8.40 (21.483)
  Change at Day 224/ET: QTcF | -4.39 (6.533) | -11.22 (11.485) | 1.94 (16.996) | 10.94 (17.055)
  Change at Day 304/ET: QTcF: number analyzed (Participants) | 0 | 6 | 6 | 4
  Change at Day 304/ET: QTcF |  | -6.72 (14.685) | -7.39 (21.754) | 11.50 (18.165)

44. Primary Outcome: Number of Participants With Positive Anti-Drug-Antibodies (ADA) and Neutralizing Antibodies (Nab)
Description: The immunogenicity of RN6G (PF-04382923) in terms of producing an antidrug antibody (ADA) and neutralizing antibody response were assessed. Neutralizing antibody response were to be assess in participants with positive ADA samples.
Time Frame: Baseline up to Day 304/ET
Population: Analysis population included all randomized participants who met the inclusion criteria and received any amount of study drug. Here "Number Analyzed" signifies number of participants evaluated for specified category. Data for Nab was not estimable as no participant was eligible for neutralizing antibody assessment, as there were no positive ADA samples.
Measure: Count of Participants; unit: Participants
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Positive ADA | 0 | 0 | 0 | 0
  Positive Nab: number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | RN6G 5 mg/kg | RN6G 10 mg/kg | RN6G 15 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RN6G 5 mg/kg (N=6) | RN6G 10 mg/kg (N=6) | RN6G 15 mg/kg (N=6) | Placebo (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RN6G 5 mg/kg (N=6) | RN6G 10 mg/kg (N=6) | RN6G 15 mg/kg (N=6) | Placebo (N=6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Age-related macular degeneration (Eye disorders) | 1 | 0 | 2 | 0
Blepharitis (Eye disorders) | 1 | 3 | 1 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 1 | 0 | 1
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Eyelid ptosis (Eye disorders) | 0 | 1 | 0 | 0
Night blindness (Eye disorders) | 0 | 0 | 1 | 0
Optic nerve sheath haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Retinal degeneration (Eye disorders) | 0 | 1 | 0 | 1
Retinal depigmentation (Eye disorders) | 0 | 1 | 0 | 0
Retinal exudates (Eye disorders) | 1 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Retinal pigmentation (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Immune system disorder (Immune system disorders) | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 4 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Venous injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Bacterial test positive (Investigations) | 2 | 0 | 0 | 0
Bilirubin urine (Investigations) | 1 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 1
Blood glucose abnormal (Investigations) | 1 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 1 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1
Complement factor C3 increased (Investigations) | 0 | 0 | 0 | 1
Complement factor increased (Investigations) | 0 | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1
Haematocrit increased (Investigations) | 1 | 0 | 0 | 0
Occult blood positive (Investigations) | 1 | 0 | 1 | 0
Optic nerve cup/disc ratio increased (Investigations) | 0 | 0 | 0 | 1
Platelet morphology abnormal (Investigations) | 1 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0
Red blood cell burr cells present (Investigations) | 1 | 0 | 0 | 0
Urinary sediment present (Investigations) | 1 | 0 | 0 | 0
Urine leukocyte esterase positive (Investigations) | 2 | 0 | 0 | 0
Visual field tests abnormal (Investigations) | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0
Cholesterosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Essential hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.